CLINICAL TRIAL: NCT05472038
Title: AN INTERVENTIONAL, RANDOMIZED, ACTIVE-CONTROLLED, PHASE 1/2/3 STUDY TO INVESTIGATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF BNT162b RNA-BASED VACCINE CANDIDATES IN COVID-19 VACCINE-EXPERIENCED HEALTHY INDIVIDUALS
Brief Title: A Study to Learn About New COVID-19 RNA Vaccine Candidates in COVID-19 Vaccine-Experienced Healthy Individuals
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C4591044; 2022-002008-19 (Registry Identifier: EudraCT); NCT05472038 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2022-07-15; First posted 2022-07-25 (Actual); Results first posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: SARS-CoV-2 Infection; COVID-19
Keywords: SARS-CoV-2 infection; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Phase 1/2/3, randomized, active-controlled, parallel group study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Cohort 1 and Cohort 2 (18 years and older): Observer-blind Cohort 2 (12-17 years) and Cohort 3: Open-label Cohort 4: Observer-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Cohort 1: BNT162b5 Bivalent (WT/OMI BA.2) (Experimental): Participants will receive 30 µg of BNT162b5 Bivalent (WT/OMI BA.2) at Visit 1.
  Interventions: Biological: BNT162b5 Bivalent (WT/OMI BA.2)
- Cohort 1: BNT162b2 Bivalent (WT/OMI BA.1) (Experimental): Participants will receive 30 µg of BNT162b2 Bivalent (WT/OMI BA.1) at Visit 1.
  Interventions: Biological: BNT162b2 Bivalent (WT/OMI BA.1)
- Cohort 2 -Group 1: 12-17 years; 30 µg (Experimental): Participants 12-17 years old will receive 30 µg of BNT162b2 Bivalent (WT/OMI BA.4/BA.5) at Visit 1.
  Interventions: Biological: BNT162b2 Bivalent (WT/OMI BA.4/BA.5)
- Cohort 2 - Group 2: 18-55 years; 30 µg (Experimental): Participants 18-55 years old will receive 30 µg of BNT162b2 Bivalent (WT/OMI BA.4/BA.5) at Visit 1.
  Interventions: Biological: BNT162b2 Bivalent (WT/OMI BA.4/BA.5)
- Cohort 2 - Group 3: 18-55 years; 60 µg (Experimental): Participants 18-55 years old will receive 60 µg of BNT162b2 Bivalent (WT/OMI BA.4/BA.5) at Visit 1.
  Interventions: Biological: BNT162b2 Bivalent (WT/OMI BA.4/BA.5)
- Cohort 2 - Group 4: >55 years; 30 µg (Experimental): Participants over 55 years old will receive 30 µg of BNT162b2 Bivalent (WT/OMI BA.4/BA.5) at Visit 1.
  Interventions: Biological: BNT162b2 Bivalent (WT/OMI BA.4/BA.5)
- Cohort 2 - Group 5: >55 years; 60 µg (Experimental): Participants over 55 years old will receive 60 µg of BNT162b2 Bivalent (WT/OMI BA.4/BA.5) at Visit 1.
  Interventions: Biological: BNT162b2 Bivalent (WT/OMI BA.4/BA.5)
- Cohort 3 - Group 1: 18-55 years; 30 µg (Experimental): Participants will receive BNT162b2 Bivalent (WT/OMI BA.4/BA.5) 30 µg at Visit 1.
  Interventions: Biological: BNT162b2 Bivalent (WT/OMI BA.4/BA.5)
- Cohort 3 - Group 2: >55 years; 30 µg (Experimental): Participants will receive BNT162b2 Bivalent (WT/OMI BA.4/BA.5) 30 µg at Visit 1.
  Interventions: Biological: BNT162b2 Bivalent (WT/OMI BA.4/BA.5)
- Cohort 4: BNT162b2 Bivalent (Original/OMI BA.4/BA.5) (Active Comparator): Participants will receive 30 µg of BNT162b2 Bivalent (Original/OMI BA.4/BA.5) at Visit 1
  Interventions: Biological: BNT162b2 Bivalent (WT/OMI BA.4/BA.5)
- Cohort 4: BNT162b5 Bivalent (Original/OMI BA.4/BA.5) (Experimental): Participants will receive 30 µg of BNT162b5 Bivalent (Original/OMI BA.4/BA.5) at Visit 1
  Interventions: Biological: BNT162b5 Bivalent (Original/OMI BA.4/BA.5)
- Cohort 4: BNT162b6 Bivalent (Original/OMI BA.4/BA.5) (Experimental): Participants will receive 30 µg of BNT162b6 Bivalent (Original/OMI BA.4/BA.5) at Visit 1
  Interventions: Biological: BNT162b6 Bivalent (Original/OMI BA.4/BA.5)
- Cohort 4: BNT162b7 Bivalent (Original/OMI BA.4/BA.5) (Experimental): Participants will receive 30 µg of BNT162b7 Bivalent (Original/OMI BA.4/BA.5) at Visit 1
  Interventions: Biological: BNT162b7 Bivalent (Original/OMI BA.4/BA.5)
- Cohort 4: BNT162b7 Monovalent (OMI BA.4/BA.5) (Experimental): Participants will receive 30 µg of BNT162b7 Monovalent (OMI BA.4/BA.5) at Visit 1
  Interventions: Biological: BNT162b7 Monovalent (OMI BA.4/BA.5)

INTERVENTIONS:
Biological: BNT162b5 Bivalent (WT/OMI BA.2) — BNT162b5 Wild Type and BNT162b5 OMICRON [B.1.1.529 sublineage BA.2]
  Arms: Cohort 1: BNT162b5 Bivalent (WT/OMI BA.2)
Biological: BNT162b2 Bivalent (WT/OMI BA.1) — BNT162b2 Wild Type and BNT162b2 OMICRON [B.1.1.529 sublineage BA.1]
  Arms: Cohort 1: BNT162b2 Bivalent (WT/OMI BA.1)
Biological: BNT162b2 Bivalent (WT/OMI BA.4/BA.5) — BNT162b2 Wild Type and BNT162b2 OMICRON [B.1.1.529 sublineage BA.4/BA.5]
  Arms: Cohort 2 - Group 2: 18-55 years; 30 µg; Cohort 2 - Group 3: 18-55 years; 60 µg; Cohort 2 - Group 4: >55 years; 30 µg; Cohort 2 - Group 5: >55 years; 60 µg; Cohort 2 -Group 1: 12-17 years; 30 µg; Cohort 3 - Group 1: 18-55 years; 30 µg; Cohort 3 - Group 2: >55 years; 30 µg; Cohort 4: BNT162b2 Bivalent (Original/OMI BA.4/BA.5)
Biological: BNT162b5 Bivalent (Original/OMI BA.4/BA.5) — BNT162b5 Wild Type and BNT162b5 OMICRON [B.1.1.529 sublineage BA.4/BA.5]
  Arms: Cohort 4: BNT162b5 Bivalent (Original/OMI BA.4/BA.5)
Biological: BNT162b6 Bivalent (Original/OMI BA.4/BA.5) — BNT162b6 Wild Type and BNT162b6 OMICRON [B.1.1.529 sublineage BA.4/BA.5]
  Arms: Cohort 4: BNT162b6 Bivalent (Original/OMI BA.4/BA.5)
Biological: BNT162b7 Bivalent (Original/OMI BA.4/BA.5) — BNT162b7 Wild Type and BNT162b7 OMICRON [B.1.1.529 sublineage BA.4/BA.5]
  Arms: Cohort 4: BNT162b7 Bivalent (Original/OMI BA.4/BA.5)
Biological: BNT162b7 Monovalent (OMI BA.4/BA.5) — BNT162b7 OMICRON [B.1.1.529 sublineage BA.4/BA.5]
  Arms: Cohort 4: BNT162b7 Monovalent (OMI BA.4/BA.5)

SUMMARY:
The purpose of this clinical trial is to learn about the safety, tolerability and immunogenicity of BNT162b RNA-based SARS-CoV-2 vaccine candidates in adults to prevent COVID-19.

For all cohorts (groups of participants), this study is seeking participants who are healthy (who may have preexisting disease if it is stable); All participants will receive a single dose of the study vaccine at the first study clinic and will return to the study clinic at least 4 more times. At each clinic visit, a blood sample will be taken. The study is about 6 months long for each participant. The vaccine candidates in this study are investigational but are very similar to BNT162b2 (Comirnaty), a COVID-19 RNA vaccine approved for use in the US and in many countries.

For Cohort 1, this study included participants who were:

* 18 through 55 years of age
* have received 1 booster dose of a US-authorized COVID-19 vaccine, with the last dose being 90 or more days before Visit 1 of this study.

All participants in Cohort 1 will receive 1 of the 2 study vaccines at a 30 microgram dose: BNT162b5 Bivalent (WT/OMI BA.2) or BNT162b2 Bivalent (WT/OMI BA.1).

For Cohort 2, this study included participants who were:

* 12 years of age and older
* have received 3 prior doses of 30 micrograms BNT162b2, with the last dose being 150 to 365 days before Visit 1 of this study.

Participants 12 through 17 years of age will receive BNT162b2 Bivalent (WT/OMI BA.4/BA.5) 30 micrograms.

Participants 18 years and older will receive BNT162b2 Bivalent (WT/OMI BA.4/BA.5) at either a 30 microgram or a 60 microgram dose.

For Cohort 3, this study included participants who were:

* 18 years of age and older
* have received 3 prior doses of 30 micrograms BNT162b2, with the last dose being 150 to 365 days before Visit 1 of this study.
* Participants will receive BNT162b2 Bivalent (WT/OMI BA.4/BA.5) 30 micrograms.

For Cohort 4, this study is seeking participants who are:

* 18 through 55 years of age
* have received 3 or 4 prior doses of a US-authorized mRNA COVID-19 vaccine (and dose level), with the last dose being a US-authorized BA.4/BA.5-adapted bivalent vaccine and dose level at least 150 days before Visit 1 of this study.

All participants in Cohort 4 will receive 1 of the 5 study vaccines at a 30 microgram dose: BNT162b2 Bivalent (Original/ OMI BA.4/BA.5), BNT162b5 Bivalent (Original/OMI BA.4/BA.5), BNT162b6 Bivalent (Original/OMI BA.4/BA.5), BNT162b7 Bivalent (Original/OMI BA.4/BA.5) or BNT162b7 Monovalent (OMI BA.4/BA.5).

ELIGIBILITY:
Inclusion Criteria:

1. Age:

   * Cohort 1: 18 through 55 years of age.
   * Cohort 2: 12 years of age and older.
   * Cohort 3: 18 years of age and older.
   * Cohort 4: 18 through 55 years of age.
2. Willing and able to comply with all scheduled visits/contacts, study procedures and lifestyle considerations.
3. Healthy participants (stable pre-existing disease permitted).
4. Capable of giving signed informed consent.
5. Prior COVID-19 vaccination history:

Cohort 1:

- Received of 1 booster dose of a US-authorized COVID-19 vaccine, with the dose being 90 or more days before first study visit. Documented receipt of all prior COVID-19 vaccines is required.

Cohorts 2 and 3:

- Received 3 prior doses of 30 micrograms BNT162b2, with last dose being 150 to 365 days before first study visit. Documented receipt of all prior COVID-19 vaccines is required.

Cohort 4:

- Received 3 or 4 prior doses of a US-authorized mRNA COVID-19 vaccine (and dose level), with the last dose being a US-authorized Omicron BA.4/BA.5-adapted vaccine and dose level at least 150 days before first study visit. Documented receipt of all prior COVID-19 vaccines is required.

Exclusion Criteria:

1. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study vaccines.
2. Known or suspected immunodeficiency.
3. Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
4. Women who are pregnant or breastfeeding.
5. Other medical or psychiatric condition, or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
6. Immunosuppressants/radiotherapy:

   Cohorts 1 and 2: Receipt of chronic systemic treatment with known immunosuppressant medications (including cytotoxic agents or systemic corticosteroids), or radiotherapy, within 60 days before study vaccination through end of study.

   Cohorts 3 and 4: Receipt of chronic systemic treatment with known immunosuppressant medications (including cytotoxic agents or systemic corticosteroids, eg, for cancer or an autoimmune disease), or radiotherapy, within 60 days before enrollment or planned receipt through conclusion of the study.
7. Blood/plasma products, immunoglobulin, or monoclonal antibodies:

   Cohorts 1, 2, 3: Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies, from 60 days before study vaccination or planned receipt throughout the study.

   Cohort 4: Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies used for treatment/prevention of COVID-19 or those considered immunosuppressive, from 60 days before study vaccination or planned receipt throughout the study.
8. Other study participation:

   Cohorts 1 and 2: Participation in other studies involving a study intervention within 28 days before randomization. Anticipated participation in other studies within 28 days after receipt of study intervention in this study.

   Cohorts 3 and 4: Participation in other studies involving receipt of a study intervention within 28 days before randomization. Anticipated participation in other studies involving a study intervention from randomization through the end of this study.
9. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.
10. Cohort 4 only: History of myocarditis or pericarditis

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1453 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (31):
- United States (31):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - California Research Foundation, San Diego, California
  - Bayview Research Group, LLC, Valley Village, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Clinical Research Consulting, Milford, Connecticut
  - Research Centers of America ( Hollywood ), Hollywood, Florida
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare, Jacksonville, Florida
  - Acevedo Clinical Research Associates, Miami, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Kentucky Pediatric/ Adult Research, Bardstown, Kentucky
  - Clinical Research Professionals, Chesterfield, Missouri
  - Sundance Clinical Research, St Louis, Missouri
  - Velocity Clinical Research, Omaha, Omaha, Nebraska
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - Rochester Clinical Research, LLC, Rochester, New York
  - Accellacare - Charlotte, Charlotte, North Carolina
  - PharmQuest Life Sciences, LLC, Greensboro, North Carolina
  - Accellacare - Wilmington, Wilmington, North Carolina
  - Senders Pediatrics, Cleveland, Ohio
  - Centricity Research Columbus Ohio Multispecialty, Columbus, Ohio
  - Kaiser Permanente Northwest Center for Health Research, Portland, Oregon
  - Clinical Neuroscience Solutions Inc., Memphis, Tennessee
  - Benchmark Research, Austin, Texas
  - Tekton Research, LLC., Austin, Texas
  - DM Clinical Research - Bellaire, Houston, Texas
  - IMA Clinical Research San Antonio, San Antonio, Texas
  - DM Clinical Research - MDC, Tomball, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - Virginia Research Center, Midlothian, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gayed J, Bangad V, Xu X, Mensa F, Cutler M, Tureci O, Sahin U, Modjarrad K, Swanson KA, Anderson AS, Gurtman A, Kitchin N; C4591054 Study Group. Immunogenicity of the Monovalent Omicron XBB.1.5-Adapted BNT162b2 COVID-19 Vaccine against XBB.1.5, BA.2.86, and JN.1 Sublineages: A Phase 2/3 Trial. Vaccines (Basel). 2024 Jul 2;12(7):734. doi: 10.3390/vaccines12070734. PMID 39066372
- [Derived] Gayed J, Diya O, Lowry FS, Xu X, Bangad V, Mensa F, Zou J, Xie X, Hu Y, Lu C, Cutler M, Belanger T, Cooper D, Koury K, Anderson AS, Tureci O, Sahin U, Swanson KA, Modjarrad K, Gurtman A, Kitchin N; C4591054 Study Group. Safety and Immunogenicity of the Monovalent Omicron XBB.1.5-Adapted BNT162b2 COVID-19 Vaccine in Individuals >/=12 Years Old: A Phase 2/3 Trial. Vaccines (Basel). 2024 Jan 24;12(2):118. doi: 10.3390/vaccines12020118. PMID 38400102
- [Derived] Usdan L, Patel S, Rodriguez H, Xu X, Lee DY, Finn D, Wyper H, Lowry FS, Mensa FJ, Lu C, Cooper D, Koury K, Anderson AS, Tureci O, Sahin U, Swanson KA, Gruber WC, Kitchin N; C4591044 Study Group. A Bivalent Omicron-BA.4/BA.5-Adapted BNT162b2 Booster in >/=12-Year-Olds. Clin Infect Dis. 2024 May 15;78(5):1194-1203. doi: 10.1093/cid/ciad718. PMID 38016021
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591044

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of 4 cohorts. Cohort 1 and 4 had distinct participant groups and objectives. Where appropriate, and as per planned analyses, data is summarized and combined for Cohort 2 (C2) and Cohort 3 (C3) 30 micrograms (mcg) groups (G) per age category to provide sufficient power for the immunogenicity hypotheses for each of the age groups.
Pre-assignment Details: Study consisted of 4 cohorts. Cohort 1 and 4 had distinct participant groups and objectives, while cohorts are different, they are part of same study. Both arms (Cohort 2 Group 2 and Cohort 3 Group 1) and (Cohort 2 Group 4 and Cohort 3 Group 2) received the same treatment and are from the same age group. As mentioned in the Protocol Objective section, arms with the same treatment and age group will be combined to provide a more comprehensive summary, rather than being listed in separate columns.
Groups:
- Cohort 1: 18-55 Years (BNT162b5 Bivalent [WT/ OMI BA.2] 30 mcg): Participants aged 18-55 years received BNT162b5 Bivalent (wild type [WT]/ omicron [OMI] BA.2) 30 micrograms (mcg) intramuscularly at Visit 1 (Day 1).
- Cohort 1: 18-55 Years (BNT162b2 Bivalent [WT/ OMI BA.1] 30 mcg): Participants aged 18-55 years received BNT162b2 Bivalent (WT/ OMI BA.1) 30 mcg intramuscularly at Visit 1 (Day 1).
- Cohort 2 (Group 1): 12-17 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 30 mcg): Participants aged 12-17 years received BNT162b2 Bivalent (WT/ OMI BA.4/ BA.5) 30 mcg intramuscularly at Visit 1 (Day 1).
- Cohort 2 (Group 2) + Cohort 3 (Group 1): 18-55 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 30 mcg): Participants aged 18-55 years received BNT162b2 Bivalent (WT/ OMI BA.4/ BA.5) 30 mcg intramuscularly at Visit 1 (Day 1).
- Cohort 2 (Group 3): 18-55 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 60 mcg): Participants aged 18-55 years received BNT162b2 Bivalent (WT/ OMI BA.4/ BA.5) 60 mcg intramuscularly at Visit 1 (Day 1).
- Cohort 2 (Group 4) + Cohort 3 (Group 2): >55 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 30 mcg): Participants aged more than (>) 55 years received BNT162b2 Bivalent (WT/ OMI BA.4/ BA.5) 30 mcg intramuscularly at Visit 1 (Day 1).
- Cohort 2 (Group 5): >55 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 60 mcg): Participants aged >55 years received BNT162b2 Bivalent (WT/ OMI BA.4/ BA.5) 60 mcg intramuscularly at Visit 1 (Day 1).
- Cohort 4: 18-55 Years (BNT162b2 Bivalent [Original/ OMI BA.4 /BA.5] 30 mcg): Participants aged 18-55 years received BNT162b2 Bivalent (Original/ OMI BA.4/ BA.5) 30 mcg intramuscularly at Visit 1 (Day 1).
- Cohort 4: 18-55 Years (BNT162b5 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg): Participants aged 18-55 years received BNT162b5 Bivalent (Original/ OMI BA.4/ BA.5) 30 mcg intramuscularly at Visit 1 (Day 1).
- Cohort 4: 18-55 Years (BNT162b6 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg): Participants aged 18-55 years received BNT162b6 Bivalent (Original/ OMI BA.4/ BA.5) 30 mcg intramuscularly at Visit 1 (Day 1).
- Cohort 4: 18-55 Years (BNT162b7 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg): Participants aged 18-55 years received BNT162b7 Bivalent (Original/ OMI BA.4/ BA.5) 30 mcg intramuscularly at Visit 1 (Day 1).
- Cohort 4: 18-55 Years (BNT162b7 Monovalent [OMI BA.4/ BA.5] 30 mcg): Participants aged 18-55 years received BNT162b7 Monovalent (OMI BA.4/ BA.5) 30 mcg intramuscularly at Visit 1 (Day 1).
Period: Overall Study
Arm/Group | Cohort 1: 18-55 Years (BNT162b5 Bivalent [WT/ OMI BA.2] 30 mcg) | Cohort 1: 18-55 Years (BNT162b2 Bivalent [WT/ OMI BA.1] 30 mcg) | Cohort 2 (Group 1): 12-17 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 30 mcg) | Cohort 2 (Group 2) + Cohort 3 (Group 1): 18-55 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 30 mcg) | Cohort 2 (Group 3): 18-55 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 60 mcg) | Cohort 2 (Group 4) + Cohort 3 (Group 2): >55 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 30 mcg) | Cohort 2 (Group 5): >55 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 60 mcg) | Cohort 4: 18-55 Years (BNT162b2 Bivalent [Original/ OMI BA.4 /BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b5 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b6 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b7 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b7 Monovalent [OMI BA.4/ BA.5] 30 mcg)
Started | 104 | 102 | 108 | 314 | 110 | 306 | 102 | 62 | 62 | 60 | 60 | 63
Completed | 102 | 96 | 103 | 298 | 106 | 300 | 101 | 59 | 57 | 58 | 55 | 59
Not Completed | 2 | 6 | 5 | 16 | 4 | 6 | 1 | 3 | 5 | 2 | 5 | 4
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 3 | 3 | 9 | 2 | 2 | 1 | 0 | 1 | 0 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 1 | 6 | 1 | 3 | 0 | 2 | 3 | 1 | 2 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1
Not completed — Not vaccinated | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study consisted of 4 cohorts. Cohort 1 and 4 had distinct participant groups and objectives, while cohorts are different, they are part of same study. Both arms (Cohort 2 Group 2 and Cohort 3 Group 1) and (Cohort 2 Group 4 and Cohort 3 Group 2) received the same treatment and are from the same age group. As mentioned in the Protocol Objective section, arms with the same treatment and age group will be combined to provide a more comprehensive summary, rather than being listed in separate columns.
Groups:
- Cohort 1: 18-55 Years (BNT162b5 Bivalent [WT/ OMI BA.2] 30 mcg): Participants aged 18-55 years received BNT162b5 Bivalent (WT/ OMI BA.2) 30 mcg intramuscularly at Visit 1 (Day 1).
- Cohort 2 (Group 4) + Cohort 3 (Group 2): >55 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 30 mcg): Participants aged > 55 years received BNT162b2 Bivalent (WT/ OMI BA.4/ BA.5) 30 mcg intramuscularly at Visit 1 (Day 1).
- Cohort 4: 18-55 Years (BNT162b2 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg): Participants aged 18-55 years received BNT162b2 Bivalent (Original/ OMI BA.4/ BA.5) 30 mcg intramuscularly at Visit 1 (Day 1).
- Total: Total of all reporting groups
Arm/Group | Cohort 1: 18-55 Years (BNT162b5 Bivalent [WT/ OMI BA.2] 30 mcg) | Cohort 1: 18-55 Years (BNT162b2 Bivalent [WT/ OMI BA.1] 30 mcg) | Cohort 2 (Group 1): 12-17 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 30 mcg) | Cohort 2 (Group 2) + Cohort 3 (Group 1): 18-55 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 30 mcg) | Cohort 2 (Group 3): 18-55 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 60 mcg) | Cohort 2 (Group 4) + Cohort 3 (Group 2): >55 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 30 mcg) | Cohort 2 (Group 5): >55 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 60 mcg) | Cohort 4: 18-55 Years (BNT162b2 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b5 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b6 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b7 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b7 Monovalent [OMI BA.4/ BA.5] 30 mcg) | Total
Number analyzed (Participants) | 104 | 102 | 108 | 314 | 110 | 306 | 102 | 62 | 62 | 60 | 60 | 63 | 1453
Age, Customized [Count of Participants; unit: Participants]
  Adolescents (12-17 years) | 0 | 0 | 108 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 108
  Adults (18-64 years) | 104 | 102 | 0 | 314 | 110 | 147 | 61 | 62 | 62 | 60 | 60 | 63 | 1145
  From 65-84 years | 0 | 0 | 0 | 0 | 0 | 157 | 40 | 0 | 0 | 0 | 0 | 0 | 197
  85 years and over | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 58 | 49 | 202 | 63 | 167 | 55 | 39 | 31 | 40 | 37 | 38 | 831
  Male | 52 | 44 | 59 | 112 | 47 | 139 | 47 | 23 | 31 | 20 | 23 | 25 | 622
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 23 | 7 | 39 | 15 | 37 | 11 | 7 | 10 | 7 | 12 | 13 | 199
  Not Hispanic or Latino | 84 | 79 | 100 | 273 | 94 | 267 | 89 | 55 | 52 | 53 | 48 | 50 | 1244
  Unknown or Not Reported | 2 | 0 | 1 | 2 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Asian | 11 | 10 | 3 | 33 | 9 | 8 | 2 | 7 | 10 | 11 | 3 | 7 | 114
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Black or African American | 10 | 15 | 9 | 26 | 11 | 48 | 8 | 4 | 11 | 6 | 3 | 4 | 155
  White | 81 | 71 | 92 | 251 | 90 | 243 | 92 | 49 | 40 | 43 | 53 | 52 | 1157
  More than one race | 1 | 4 | 3 | 4 | 0 | 3 | 0 | 2 | 1 | 0 | 0 | 0 | 18
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Percentage of Participants Reporting Local Reactions Within 7 Days After Study Vaccination
Description: Local reactions were recorded by participants in an electronic diary (e-diary). Local reactions included redness, swelling and pain at injection site. Redness and swelling were graded as mild: greater than (>) 2.0 to 5.0 centimeter (cm), moderate: >5.0 to 10.0 cm, severe: >10.0 cm, grade 4 (potentially life threatening): necrosis or exfoliative dermatitis (redness) and necrosis (swelling). Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfered with daily activity, severe: prevented daily activity and grade 4 (potentially life threatening): emergency room visit or hospitalization for severe pain. Grade 4 reactions were classified by the investigator or medically qualified person. Local reactions reported as adverse events (AEs) in the case report form within 7 days after the study vaccination were also reported.
Time Frame: From Day 1 to Day 7 after study vaccination
Population: Safety population included all participants who received the study intervention and where appropriate informed consent was obtained.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Cohort 1: 18-55 Years (BNT162b5 Bivalent [WT/OMI BA.2] 30 mcg): Participants aged 18-55 years received BNT162b5 Bivalent (WT/OMI] BA.2) 30 mcg intramuscularly at Visit 1 (Day 1).
- Cohort 1: 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.1] 30 mcg): Participants aged 18-55 years received BNT162b2 Bivalent (WT/OMI BA.1) 30 mcg intramuscularly at Visit 1 (Day 1).
Arm/Group | Cohort 1: 18-55 Years (BNT162b5 Bivalent [WT/OMI BA.2] 30 mcg) | Cohort 1: 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.1] 30 mcg)
Number analyzed (Participants) | 104 | 102
Percentage of participants
  Redness: Any | 5.8 [2.1 to 12.1] | 5.9 [2.2 to 12.4]
  Redness: Mild | 3.8 [1.1 to 9.6] | 3.9 [1.1 to 9.7]
  Redness: Moderate | 1.0 [0.0 to 5.2] | 2.0 [0.2 to 6.9]
  Redness: Severe | 1.0 [0.0 to 5.2] | 0 [0.0 to 3.6]
  Redness: Grade 4 | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  Swelling: Any | 10.6 [5.4 to 18.1] | 10.8 [5.5 to 18.5]
  Swelling: Mild | 6.7 [2.7 to 13.4] | 4.9 [1.6 to 11.1]
  Swelling: Moderate | 2.9 [0.6 to 8.2] | 5.9 [2.2 to 12.4]
  Swelling: Severe | 1.0 [0.0 to 5.2] | 0 [0.0 to 3.6]
  Swelling: Grade 4 | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  Pain at injection site: Any | 82.7 [74.0 to 89.4] | 81.4 [72.4 to 88.4]
  Pain at injection site: Mild | 67.3 [57.4 to 76.2] | 62.7 [52.6 to 72.1]
  Pain at injection site: Moderate | 15.4 [9.1 to 23.8] | 18.6 [11.6 to 27.6]
  Pain at injection site: Severe | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  Pain at injection site: Grade 4 | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]

2. Primary Outcome: Cohort 1: Percentage of Participants Reporting Systemic Events Within 7 Days After Study Vaccination
Description: Systemic events were recorded by participants in an e-diary. Fever was oral temperature greater than or equal to (>=) 38 degree Celsius (deg C) and categorized as >=38.0 to 38.4 deg C, >38.4 to 38.9 deg C, >38.9 to 40.0 deg C and >40.0 deg C. Fatigue, headache, chills, new or worsened muscle pain and new or worsened joint pain were graded as mild: did not interfere with activity, moderate: some interference with activity and severe: prevented daily routine activity. Vomiting was graded as mild: 1 to 2 times in 24 hours (h), moderate: >2 times in 24h and severe: required intravenous hydration. Diarrhea was graded as mild: 2 to 3 loose stools in 24h, moderate: 4 to 5 loose stools in 24h and severe: 6 or more loose stools in 24h. For all systemic events except fever, Grade 4= emergency room visit or hospitalization. Grade 4 events were classified by the investigator/medically qualified person. Systemic events reported as AEs in the CRF within 7 days after vaccination were also reported.
Time Frame: From Day 1 to Day 7 after study vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Cohort 1: 18-55 Years (BNT162b5 Bivalent [WT/OMI BA.2] 30 mcg): Participants aged 18-55 years received BNT162b5 Bivalent (WT/OMI BA.2) 30 mcg intramuscularly at Visit 1 (Day 1).
Arm/Group | Cohort 1: 18-55 Years (BNT162b5 Bivalent [WT/OMI BA.2] 30 mcg) | Cohort 1: 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.1] 30 mcg)
Number analyzed (Participants) | 104 | 102
Percentage of participants
  Fever: Any | 1.9 [0.2 to 6.8] | 5.9 [2.2 to 12.4]
  Fever: >=38.0 deg C to 38.4 deg C | 1.0 [0.0 to 5.2] | 2.0 [0.2 to 6.9]
  Fever: >38.4 deg C to 38.9 deg C | 0 [0.0 to 3.5] | 1.0 [0.0 to 5.3]
  Fever: >38.9 deg C to 40.0 deg C | 1.0 [0.0 to 5.2] | 2.9 [0.6 to 8.4]
  Fever: >40.0 deg C | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  Fatigue: Any | 73.1 [63.5 to 81.3] | 62.7 [52.6 to 72.1]
  Fatigue: Mild | 37.5 [28.2 to 47.5] | 27.5 [19.1 to 37.2]
  Fatigue: Moderate | 34.6 [25.6 to 44.6] | 34.3 [25.2 to 44.4]
  Fatigue: Severe | 1.0 [0.0 to 5.2] | 1.0 [0.0 to 5.3]
  Fatigue: Grade 4 | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  Headache: Any | 52.9 [42.8 to 62.8] | 46.1 [36.2 to 56.2]
  Headache: Mild | 29.8 [21.2 to 39.6] | 22.5 [14.9 to 31.9]
  Headache: Moderate | 21.2 [13.8 to 30.3] | 22.5 [14.9 to 31.9]
  Headache: Severe | 1.9 [0.2 to 6.8] | 1.0 [0.0 to 5.3]
  Headache: Grade 4 | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  Chills: Any | 21.2 [13.8 to 30.3] | 19.6 [12.4 to 28.6]
  Chills: Mild | 10.6 [5.4 to 18.1] | 7.8 [3.4 to 14.9]
  Chills: Moderate | 10.6 [5.4 to 18.1] | 11.8 [6.2 to 19.6]
  Chills: Severe | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  Chills: Grade 4 | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  Vomiting: Any | 1.0 [0.0 to 5.2] | 2.0 [0.2 to 6.9]
  Vomiting: Mild | 1.0 [0.0 to 5.2] | 2.0 [0.2 to 6.9]
  Vomiting: Moderate | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  Vomiting: Severe | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  Vomiting: Grade 4 | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  Diarrhea: Any | 14.4 [8.3 to 22.7] | 19.6 [12.4 to 28.6]
  Diarrhea: Mild | 13.5 [7.6 to 21.6] | 14.7 [8.5 to 23.1]
  Diarrhea: Moderate | 1.0 [0.0 to 5.2] | 3.9 [1.1 to 9.7]
  Diarrhea: Severe | 0 [0.0 to 3.5] | 1.0 [0.0 to 5.3]
  Diarrhea: Grade 4 | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  New or worsened muscle pain: Any | 35.6 [26.4 to 45.6] | 38.2 [28.8 to 48.4]
  New or worsened muscle pain: Mild | 18.3 [11.4 to 27.1] | 23.5 [15.7 to 33.0]
  New or worsened muscle pain: Moderate | 17.3 [10.6 to 26.0] | 14.7 [8.5 to 23.1]
  New or worsened muscle pain: Severe | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  New or worsened muscle pain: Grade 4 | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  New or worsened joint pain: Any | 18.3 [11.4 to 27.1] | 17.6 [10.8 to 26.4]
  New or worsened joint pain: Mild | 7.7 [3.4 to 14.6] | 11.8 [6.2 to 19.6]
  New or worsened joint pain: Moderate | 10.6 [5.4 to 18.1] | 5.9 [2.2 to 12.4]
  New or worsened joint pain: Severe | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  New or worsened joint pain: Grade 4 | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]

3. Primary Outcome: Cohort 1: Percentage of Participants With Adverse Events (AEs) From Study Vaccination Through 1 Month After Study Vaccination
Description: An AE was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. Results excluded local reactions and systemic events data.
Time Frame: From study vaccination on Day 1 through 1 month after study vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: 18-55 Years (BNT162b5 Bivalent [WT/OMI BA.2] 30 mcg) | Cohort 1: 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.1] 30 mcg)
Number analyzed (Participants) | 104 | 102
Percentage of participants | 8.7 [4.0 to 15.8] | 12.7 [7.0 to 20.8]

4. Primary Outcome: Cohort 1: Percentage of Participants With Serious Adverse Events (SAEs) From Study Vaccination Through 6 Months After Study Vaccination
Description: An AE was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was an AE that resulted in death, was life-threatening, resulted in persistent disability/incapacity; constituted a congenital anomaly/birth defect; was important medical event, medical event was judged by investigator; required inpatient hospitalization or prolongation of existing hospitalization.
Time Frame: From study vaccination on Day 1 through 6 months after study vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Cohort 1: 18-55 Years (BNT162b5 Bivalent [WT/OMI BA.2] 30 mcg: Participants aged 18-55 years received BNT162b5 Bivalent (WT/OMI BA.2) 30 mcg intramuscularly at Visit 1 (Day 1).
Arm/Group | Cohort 1: 18-55 Years (BNT162b5 Bivalent [WT/OMI BA.2] 30 mcg | Cohort 1: 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.1] 30 mcg)
Number analyzed (Participants) | 104 | 102
Percentage of participants | 1.0 [0.0 to 5.2] | 2.0 [0.2 to 6.9]

5. Primary Outcome: Cohort 1: Geometric Mean Titer (GMT) of SARS-CoV-2 Omicron Strain (BA.1 and BA.2) and Reference Strain Neutralizing Titers (NTs) at Baseline- Participants Without Evidence of Infection
Description: GMTs and the corresponding 2-sided confidence intervals (CIs) were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on student's t distribution). Assay results below the lower limit of quantification (LLOQ) were set to 0.5*LLOQ.
Time Frame: At baseline (before study vaccination)
Population: Evaluable immunogenicity population (EIP): randomized participants who received intervention to which they were randomized, 1 valid, determinate immunogenicity result from blood sample collected 28-42 days post vaccination, no important protocol deviations. Analysis performed in participants without evidence of infection up to 1 month post vaccination. Overall Number of Participants Analyzed= participants evaluable for outcome measure; Number Analyzed= participants evaluable for specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 1: 18-55 Years (BNT162b5 Bivalent [WT/OMI BA.2] 30 mcg) | Cohort 1: 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.1] 30 mcg)
Number analyzed (Participants) | 30 | 29
Titer
  Omicron BA.2: number analyzed (Participants) | 29 | 29
  Omicron BA.2 | 169.3 [96.7 to 296.3] | 377.8 [229.2 to 622.8]
  Omicron BA.1 | 103.3 [60.4 to 176.6] | 209.5 [147.2 to 298.2]
  Reference strain | 892.0 [526.5 to 1511.3] | 1544.2 [993.8 to 2399.4]

6. Primary Outcome: Cohort 1: GMT of SARS-CoV-2 Omicron Strain (BA.1 and BA.2) and Reference Strain NTs at Baseline- Participants With or Without Evidence of Infection
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on student's t distribution).
Time Frame: At baseline (before study vaccination)
Population: EIP: all eligible randomized/assigned participants who received study intervention to which they were randomized/assigned, had at least 1 valid, determinate immunogenicity result from blood sample collected within 28-42 days after study vaccination, had no other important protocol deviations as determined by clinician. Analysis was performed in participants with or without evidence of infection up to 1 month post study vaccination. ''Number Analyzed'' =participants evaluable for specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 1: 18-55 Years (BNT162b5 Bivalent [WT/OMI BA.2] 30 mcg) | Cohort 1: 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.1] 30 mcg)
Number analyzed (Participants) | 103 | 98
Titer
  Omicron BA.2: number analyzed (Participants) | 102 | 96
  Omicron BA.2 | 1269.1 [854.7 to 1884.6] | 1527.5 [1061.3 to 2198.6]
  Omicron BA.1 | 652.7 [448.9 to 949.0] | 818.7 [595.9 to 1124.7]
  Reference strain | 3469.8 [2536.5 to 4746.7] | 3755.9 [2896.8 to 4869.9]

7. Primary Outcome: Cohort 1: GMT of SARS-CoV-2 Omicron Strain (BA.1 and BA.2) and Reference Strain NTs at 1 Month After Study Vaccination- Participants Without Evidence of Infection
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on student's t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: 1 month after the study vaccination
Population: EIP: randomized participants who received intervention to which they were randomized, 1 valid, determinate immunogenicity result from blood sample collected 28-42 days post vaccination, no important protocol deviations. Analysis performed in participants without evidence of infection up to 1 month post vaccination. Here, ''Overall Number of Participants Analyzed'' signifies participants evaluable for this outcome measure; ''Number Analyzed'' signifies participants evaluable for specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 1: 18-55 Years (BNT162b5 Bivalent [WT/OMI BA.2] 30 mcg) | Cohort 1: 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.1] 30 mcg)
Number analyzed (Participants) | 30 | 29
Titer
  Omicron BA.2: number analyzed (Participants) | 30 | 28
  Omicron BA.2 | 2414.8 [1508.5 to 3865.4] | 2768.5 [1948.5 to 3933.7]
  Omicron BA.1 | 1666.1 [1085.8 to 2556.6] | 1993.8 [1309.1 to 3036.6]
  Reference strain | 8268.9 [5901.9 to 11585.1] | 7391.6 [5117.5 to 10676.2]

8. Primary Outcome: Cohort 1: GMT of SARS-CoV-2 Omicron Strain (BA.1 and BA.2) and Reference Strain NTs at 1 Month After Study Vaccination- Participants With or Without Evidence of Infection
Description: as for outcome 7
Time Frame: 1 month after the study vaccination
Population: EIP: all eligible randomized/assigned participants who received study intervention to which they were randomized/assigned, had at least 1 valid, determinate immunogenicity result from blood sample collected within 28-42 days after study vaccination, had no other important protocol deviations as determined by clinician. Analysis was performed in participants with or without evidence of infection up to 1 month post study vaccination. ''Number Analyzed'' = participants evaluable for specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 1: 18-55 Years (BNT162b5 Bivalent [WT/OMI BA.2] 30 mcg) | Cohort 1: 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.1] 30 mcg)
Number analyzed (Participants) | 103 | 98
Titer
  Omicron BA.2: number analyzed (Participants) | 102 | 95
  Omicron BA.2 | 6267.9 [4766.0 to 8243.1] | 4984.2 [3976.4 to 6247.4]
  Omicron BA.1 | 3582.2 [2813.7 to 4560.7] | 3571.8 [2899.6 to 4399.8]
  Reference strain | 14342.3 [11811.9 to 17414.9] | 11246.8 [9395.1 to 13463.6]

9. Primary Outcome: Cohort 1: Geometric Mean Fold Rise (GMFR) of SARS-CoV-2 Omicron Strain (BA.1 and BA.2) and Reference Strain- NTs From Before the Study Vaccination to 1 Month After the Study Vaccination- Participants Without Evidence of Infection
Description: GMFR from before study vaccination to 1 month after study vaccination for each strain-specific neutralizing titer was reported in this endpoint. GMFRs and 2-sided 95% CIs were calculated by exponentiating mean logarithm of fold rises and corresponding CIs (based on student-t distribution). Assay results below lower limit of quantitation (LLOQ) were set to 0.5*LLOQ in analysis.
Time Frame: From before the study vaccination to 1 month after the study vaccination
Population: as for outcome 7
Measure: Geometric Mean (96% Confidence Interval); unit: Fold rise
Arm/Group | Cohort 1: 18-55 Years (BNT162b5 Bivalent [WT/OMI BA.2] 30 mcg) | Cohort 1: 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.1] 30 mcg)
Number analyzed (Participants) | 30 | 29
Fold rise
  Omicron BA.2: number analyzed (Participants) | 29 | 28
  Omicron BA.2 | 14.6 [8.4 to 25.5] | 6.9 [4.4 to 10.9]
  Omicron BA.1 | 16.1 [10.9 to 23.9] | 9.5 [6.5 to 13.8]
  Reference strain | 9.3 [5.9 to 14.6] | 4.8 [3.1 to 7.3]

10. Primary Outcome: Cohort 1: GMFR of SARS-CoV-2 Omicron Strain (BA.1 and BA2) and Reference Strain- NTs From Before the Study Vaccination to 1 Month After the Study Vaccination- Participants With or Without Evidence of Infection
Description: GMFR from before study vaccination to 1 month after study vaccination for each strain-specific neutralizing titer was reported in this endpoint. GMFRs and 2-sided 95% CIs were calculated by exponentiating mean logarithm of fold rises and corresponding CIs (based on student-t distribution). Assay results below LLOQ were set to 0.5*LLOQ in analysis.
Time Frame: From before the study vaccination to 1 month after the study vaccination
Population: EIP: all eligible randomized/assigned participants who received study intervention to which they were randomized/assigned, had at least 1 valid, determinate immunogenicity result from blood sample collected within 28-42 days after study vaccination, had no other important protocol deviations as determined by clinician. Analysis was performed in participants with or without evidence of infection up to 1 month post study vaccination. ''Number Analyzed''= participants evaluable for specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Cohort 1: 18-55 Years (BNT162b5 Bivalent [WT/OMI BA.2] 30 mcg) | Cohort 1: 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.1] 30 mcg)
Number analyzed (Participants) | 103 | 98
Fold rise
  Omicron BA.2: number analyzed (Participants) | 101 | 93
  Omicron BA.2 | 5.0 [3.6 to 6.8] | 3.2 [2.3 to 4.3]
  Omicron BA.1 | 5.5 [4.3 to 7.1] | 4.4 [3.4 to 5.6]
  Reference strain | 4.1 [3.3 to 5.2] | 3.0 [2.4 to 3.7]

11. Primary Outcome: Cohort 1: Percentage of Participants With Seroresponse to SARS-CoV-2 Omicron Strain (BA.1 and BA.2) and Reference Strain- NTs at 1 Month After Study Vaccination- Participants Without Evidence of Infection
Description: Seroresponse was defined as achieving >= 4-fold rise in NTs from baseline (before the study vaccination). If the baseline measurement was below the LLOQ, the postvaccination measure of >= 4*LLOQ was considered a seroresponse.
Time Frame: 1 month after the study vaccination
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: 18-55 Years (BNT162b5 Bivalent [WT/OMI BA.2] 30 mcg) | Cohort 1: 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.1] 30 mcg)
Number analyzed (Participants) | 30 | 29
Percentage of participants
  Omicron BA.2: number analyzed (Participants) | 29 | 28
  Omicron BA.2 | 82.8 [64.2 to 94.2] | 71.4 [51.3 to 86.8]
  Omicron BA.1 | 93.3 [77.9 to 99.2] | 86.2 [68.3 to 96.1]
  Reference strain | 73.3 [54.1 to 87.7] | 51.7 [32.5 to 70.6]

12. Primary Outcome: Cohort 1: Percentage of Participants With Seroresponse to SARS-CoV-2 Omicron Strain (BA.1 and BA.2) and Reference Strain- NTs at 1 Month After Study Vaccination- Participants With or Without Evidence of Infection
Description: as for outcome 11
Time Frame: 1 month after the study vaccination
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: 18-55 Years (BNT162b5 Bivalent [WT/OMI BA.2] 30 mcg) | Cohort 1: 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.1] 30 mcg)
Number analyzed (Participants) | 103 | 98
Percentage of participants
  Omicron BA.2: number analyzed (Participants) | 101 | 93
  Omicron BA.2 | 53.5 [43.3 to 63.5] | 40.9 [30.8 to 51.5]
  Omicron BA.1 | 58.3 [48.1 to 67.9] | 49.0 [38.7 to 59.3]
  Reference strain | 43.7 [33.9 to 53.8] | 30.6 [21.7 to 40.7]

13. Primary Outcome: Cohort 2: Percentage of Participants Reporting Local Reactions Within 7 Days After Study Vaccination
Description: Local reactions were recorded by participants in an e-diary. Local reactions included redness, swelling and pain at injection site. Redness and swelling were graded as mild: > 2.0 to 5.0 cm, moderate: >5.0 to 10.0 cm, severe: >10.0 cm, grade 4 (potentially life threatening): necrosis or exfoliative dermatitis (redness) and necrosis (swelling). Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfered with daily activity, severe: prevented daily activity and grade 4 (potentially life threatening): emergency room visit or hospitalization for severe pain. Grade 4 reactions were classified by the investigator or medically qualified person. Local reactions reported as AEs in the case report form within 7 days after the study vaccination were also reported.
Time Frame: From Day 1 to Day 7 after study vaccination
Population: Safety population included all participants who received the study intervention and where appropriate informed consent was obtained. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and ''Number Analyzed'' signifies participants evaluable for the specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Cohort 2 (Group 1): 12-17 Years (BNT162b2 [WT/OMI BA.4/BA.5] 30 mcg): Participants aged 12-17 years received BNT162b2 Bivalent (WT/OMI BA.4/BA.5) 30 mcg intramuscularly at Visit 1 (Day 1).
- Cohort 2 (Group 2): 18-55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 30 mcg): Participants aged 18-55 years received BNT162b2 Bivalent (WT/OMI BA.4/BA.5) 30 mcg intramuscularly at Visit 1 (Day 1).
- Cohort 2 (Group 3): 18-55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 60 mcg): Participants aged 18-55 years received BNT162b2 Bivalent (WT/OMI BA.4/BA.5) 60 mcg intramuscularly at Visit 1 (Day 1).
- Cohort 2 (Group 4): >55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 30 mcg): Participants aged >55 years received BNT162b2 Bivalent (WT/OMI BA.4/BA.5) 30 mcg intramuscularly at Visit 1 (Day 1).
- Cohort 2 (Group 5): >55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 60 mcg): Participants aged >55 years received BNT162b2 Bivalent (WT/OMI BA.4/BA.5) 60 mcg intramuscularly at Visit 1 (Day 1).
Arm/Group | Cohort 2 (Group 1): 12-17 Years (BNT162b2 [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 2): 18-55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 3): 18-55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 60 mcg) | Cohort 2 (Group 4): >55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 5): >55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 60 mcg)
Number analyzed (Participants) | 107 | 102 | 110 | 105 | 102
Percentage of participants
  Redness: Any: number analyzed (Participants) | 107 | 102 | 110 | 105 | 101
  Redness: Any | 5.6 [2.1 to 11.8] | 5.9 [2.2 to 12.4] | 10.9 [5.8 to 18.3] | 2.9 [0.6 to 8.1] | 6.9 [2.8 to 13.8]
  Redness: Mild: number analyzed (Participants) | 107 | 102 | 110 | 105 | 101
  Redness: Mild | 3.7 [1.0 to 9.3] | 4.9 [1.6 to 11.1] | 5.5 [2.0 to 11.5] | 1.0 [0.0 to 5.2] | 4.0 [1.1 to 9.8]
  Redness: Moderate: number analyzed (Participants) | 107 | 102 | 110 | 105 | 101
  Redness: Moderate | 1.9 [0.2 to 6.6] | 1.0 [0.0 to 5.3] | 4.5 [1.5 to 10.3] | 1.9 [0.2 to 6.7] | 3.0 [0.6 to 8.4]
  Redness: Severe: number analyzed (Participants) | 107 | 102 | 110 | 105 | 101
  Redness: Severe | 0 [0.0 to 3.4] | 0 [0.0 to 3.6] | 0.9 [0.0 to 5.0] | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  Redness: Grade 4: number analyzed (Participants) | 107 | 102 | 110 | 105 | 101
  Redness: Grade 4 | 0 [0.0 to 3.4] | 0 [0.0 to 3.6] | 0 [0.0 to 3.3] | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  Swelling: Any: number analyzed (Participants) | 107 | 102 | 110 | 105 | 101
  Swelling: Any | 7.5 [3.3 to 14.2] | 6.9 [2.8 to 13.6] | 15.5 [9.3 to 23.6] | 1.9 [0.2 to 6.7] | 8.9 [4.2 to 16.2]
  Swelling: Mild: number analyzed (Participants) | 107 | 102 | 110 | 105 | 101
  Swelling: Mild | 5.6 [2.1 to 11.8] | 4.9 [1.6 to 11.1] | 6.4 [2.6 to 12.7] | 1.0 [0.0 to 5.2] | 5.0 [1.6 to 11.2]
  Swelling: Moderate: number analyzed (Participants) | 107 | 102 | 110 | 105 | 101
  Swelling: Moderate | 1.9 [0.2 to 6.6] | 2.0 [0.2 to 6.9] | 9.1 [4.4 to 16.1] | 1.0 [0.0 to 5.2] | 4.0 [1.1 to 9.8]
  Swelling: Severe: number analyzed (Participants) | 107 | 102 | 110 | 105 | 101
  Swelling: Severe | 0 [0.0 to 3.4] | 0 [0.0 to 3.6] | 0 [0.0 to 3.3] | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  Swelling: Grade 4: number analyzed (Participants) | 107 | 102 | 110 | 105 | 101
  Swelling: Grade 4 | 0 [0.0 to 3.4] | 0 [0.0 to 3.6] | 0 [0.0 to 3.3] | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  Pain at the injection site: Any | 70.1 [60.5 to 78.6] | 79.4 [70.3 to 86.8] | 93.6 [87.3 to 97.4] | 56.2 [46.2 to 65.9] | 70.6 [60.7 to 79.2]
  Pain at the injection site: Mild | 42.1 [32.6 to 52.0] | 63.7 [53.6 to 73.0] | 53.6 [43.9 to 63.2] | 50.5 [40.5 to 60.4] | 52.9 [42.8 to 62.9]
  Pain at the injection site: Moderate | 27.1 [19.0 to 36.6] | 15.7 [9.2 to 24.2] | 40.0 [30.8 to 49.8] | 5.7 [2.1 to 12.0] | 17.6 [10.8 to 26.4]
  Pain at the injection site: Severe | 0.9 [0.0 to 5.1] | 0 [0.0 to 3.6] | 0 [0.0 to 3.3] | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  Pain at the injection site: Grade 4 | 0 [0.0 to 3.4] | 0 [0.0 to 3.6] | 0 [0.0 to 3.3] | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]

14. Primary Outcome: Cohort 2: Percentage of Participants Reporting Systemic Events Within 7 Days After Study Vaccination
Description: Systemic events were recorded by participants in an e-diary. Fever was oral temperature >= 38 deg C and categorized as >=38.0 to 38.4 deg C, >38.4 to 38.9 deg C, >38.9 to 40.0 deg C and >40.0 deg C. Fatigue, headache, chills, new or worsened muscle pain and new or worsened joint pain were graded as mild: did not interfere with activity, moderate: some interference with activity and severe: prevented daily routine activity. Vomiting was graded as mild: 1 to 2 times in 24h, moderate: >2 times in 24h and severe: required intravenous hydration. Diarrhea was graded as mild: 2 to 3 loose stools in 24h, moderate: 4 to 5 loose stools in 24h and severe: 6 or more loose stools in 24h. For all systemic events except fever, Grade 4= emergency room visit or hospitalization. Grade 4 events were classified by the investigator or medically qualified person. Systemic events reported as AEs in the CRF within 7 days after vaccination were also reported.
Time Frame: From Day 1 to Day 7 after study vaccination
Population: Safety population included all participants who received the study intervention and where appropriate informed consent was obtained. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2 (Group 1): 12-17 Years (BNT162b2 [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 2): 18-55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 3): 18-55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 60 mcg) | Cohort 2 (Group 4): >55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 5): >55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 60 mcg)
Number analyzed (Participants) | 107 | 102 | 110 | 105 | 101
Percentage of participants
  Fever: Any | 9.3 [4.6 to 16.5] | 4.9 [1.6 to 11.1] | 11.8 [6.4 to 19.4] | 7.6 [3.3 to 14.5] | 13.9 [7.8 to 22.2]
  Fever: >=38.0 deg C to 38.4 deg C | 6.5 [2.7 to 13.0] | 2.0 [0.2 to 6.9] | 7.3 [3.2 to 13.8] | 5.7 [2.1 to 12.0] | 7.9 [3.5 to 15.0]
  Fever: >38.4 deg C to 38.9 deg C | 1.9 [0.2 to 6.6] | 2.9 [0.6 to 8.4] | 2.7 [0.6 to 7.8] | 1.9 [0.2 to 6.7] | 4.0 [1.1 to 9.8]
  Fever: >38.9 deg C to 40.0 deg C | 0.9 [0.0 to 5.1] | 0 [0.0 to 3.6] | 1.8 [0.2 to 6.4] | 0 [0.0 to 3.5] | 2.0 [0.2 to 7.0]
  Fever: >40.0 deg C | 0 [0.0 to 3.4] | 0 [0.0 to 3.6] | 0 [0.0 to 3.3] | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  Fatigue: Any | 67.3 [57.5 to 76.0] | 62.7 [52.6 to 72.1] | 69.1 [59.6 to 77.6] | 39.0 [29.7 to 49.1] | 53.5 [43.3 to 63.5]
  Fatigue: Mild | 25.2 [17.3 to 34.6] | 30.4 [21.7 to 40.3] | 24.5 [16.8 to 33.7] | 20.0 [12.8 to 28.9] | 23.8 [15.9 to 33.3]
  Fatigue: Moderate | 42.1 [32.6 to 52.0] | 30.4 [21.7 to 40.3] | 43.6 [34.2 to 53.4] | 18.1 [11.3 to 26.8] | 25.7 [17.6 to 35.4]
  Fatigue: Severe | 0 [0.0 to 3.4] | 2.0 [0.2 to 6.9] | 0.9 [0.0 to 5.0] | 1.0 [0.0 to 5.2] | 4.0 [1.1 to 9.8]
  Fatigue: Grade 4 | 0 [0.0 to 3.4] | 0 [0.0 to 3.6] | 0 [0.0 to 3.3] | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  Headache: Any | 50.5 [40.6 to 60.3] | 44.1 [34.3 to 54.3] | 45.5 [35.9 to 55.2] | 29.5 [21.0 to 39.2] | 35.6 [26.4 to 45.8]
  Headache: Mild | 26.2 [18.1 to 35.6] | 32.4 [23.4 to 42.3] | 27.3 [19.2 to 36.6] | 21.9 [14.4 to 31.0] | 20.8 [13.4 to 30.0]
  Headache: Moderate | 24.3 [16.5 to 33.5] | 11.8 [6.2 to 19.6] | 17.3 [10.7 to 25.7] | 7.6 [3.3 to 14.5] | 13.9 [7.8 to 22.2]
  Headache: Severe | 0 [0.0 to 3.4] | 0 [0.0 to 3.6] | 0.9 [0.0 to 5.0] | 0 [0.0 to 3.5] | 1.0 [0.0 to 5.4]
  Headache: Grade 4 | 0 [0.0 to 3.4] | 0 [0.0 to 3.6] | 0 [0.0 to 3.3] | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  Chills: Any | 23.4 [15.7 to 32.5] | 14.7 [8.5 to 23.1] | 27.3 [19.2 to 36.6] | 12.4 [6.8 to 20.2] | 22.8 [15.0 to 32.2]
  Chills: Mild | 17.8 [11.0 to 26.3] | 8.8 [4.1 to 16.1] | 17.3 [10.7 to 25.7] | 6.7 [2.7 to 13.3] | 11.9 [6.3 to 19.8]
  Chills: Moderate | 5.6 [2.1 to 11.8] | 5.9 [2.2 to 12.4] | 9.1 [4.4 to 16.1] | 5.7 [2.1 to 12.0] | 10.9 [5.6 to 18.7]
  Chills: Severe | 0 [0.0 to 3.4] | 0 [0.0 to 3.6] | 0.9 [0.0 to 5.0] | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  Chills: Grade 4 | 0 [0.0 to 3.4] | 0 [0.0 to 3.6] | 0 [0.0 to 3.3] | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  Vomiting: Any | 2.8 [0.6 to 8.0] | 2.0 [0.2 to 6.9] | 1.8 [0.2 to 6.4] | 1.0 [0.0 to 5.2] | 3.0 [0.6 to 8.4]
  Vomiting: Mild | 2.8 [0.6 to 8.0] | 1.0 [0.0 to 5.3] | 0.9 [0.0 to 5.0] | 1.0 [0.0 to 5.2] | 2.0 [0.2 to 7.0]
  Vomiting: Moderate | 0 [0.0 to 3.4] | 1.0 [0.0 to 5.3] | 0.9 [0.0 to 5.0] | 0 [0.0 to 3.5] | 1.0 [0.0 to 5.4]
  Vomiting: Severe | 0 [0.0 to 3.4] | 0 [0.0 to 3.6] | 0 [0.0 to 3.3] | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  Vomiting: Grade 4 | 0 [0.0 to 3.4] | 0 [0.0 to 3.6] | 0 [0.0 to 3.3] | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  Diarrhea: Any | 6.5 [2.7 to 13.0] | 13.7 [7.7 to 22.0] | 12.7 [7.1 to 20.4] | 8.6 [4.0 to 15.6] | 6.9 [2.8 to 13.8]
  Diarrhea: Mild | 6.5 [2.7 to 13.0] | 9.8 [4.8 to 17.3] | 11.8 [6.4 to 19.4] | 8.6 [4.0 to 15.6] | 5.9 [2.2 to 12.5]
  Diarrhea: Moderate | 0 [0.0 to 3.4] | 2.9 [0.6 to 8.4] | 0.9 [0.0 to 5.0] | 0 [0.0 to 3.5] | 1.0 [0.0 to 5.4]
  Diarrhea: Severe | 0 [0.0 to 3.4] | 1.0 [0.0 to 5.3] | 0 [0.0 to 3.3] | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  Diarrhea: Grade 4 | 0 [0.0 to 3.4] | 0 [0.0 to 3.6] | 0 [0.0 to 3.3] | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  New or worsened muscle pain: Any | 26.2 [18.1 to 35.6] | 31.4 [22.5 to 41.3] | 41.8 [32.5 to 51.6] | 20.0 [12.8 to 28.9] | 22.8 [15.0 to 32.2]
  New or worsened muscle pain: Mild | 11.2 [5.9 to 18.8] | 17.6 [10.8 to 26.4] | 21.8 [14.5 to 30.7] | 12.4 [6.8 to 20.2] | 12.9 [7.0 to 21.0]
  New or worsened muscle pain: Moderate | 15.0 [8.8 to 23.1] | 13.7 [7.7 to 22.0] | 19.1 [12.2 to 27.7] | 7.6 [3.3 to 14.5] | 8.9 [4.2 to 16.2]
  New or worsened muscle pain: Severe | 0 [0.0 to 3.4] | 0 [0.0 to 3.6] | 0.9 [0.0 to 5.0] | 0 [0.0 to 3.5] | 1.0 [0.0 to 5.4]
  New or worsened muscle pain: Grade 4 | 0 [0.0 to 3.4] | 0 [0.0 to 3.6] | 0 [0.0 to 3.3] | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]
  New or worsened joint pain: Any | 12.1 [6.6 to 19.9] | 16.7 [10.0 to 25.3] | 24.5 [16.8 to 33.7] | 11.4 [6.0 to 19.1] | 14.9 [8.6 to 23.3]
  New or worsened joint pain: Mild | 8.4 [3.9 to 15.4] | 9.8 [4.8 to 17.3] | 11.8 [6.4 to 19.4] | 6.7 [2.7 to 13.3] | 5.9 [2.2 to 12.5]
  New or worsened joint pain: Moderate | 3.7 [1.0 to 9.3] | 6.9 [2.8 to 13.6] | 11.8 [6.4 to 19.4] | 4.8 [1.6 to 10.8] | 7.9 [3.5 to 15.0]
  New or worsened joint pain: Severe | 0 [0.0 to 3.4] | 0 [0.0 to 3.6] | 0.9 [0.0 to 5.0] | 0 [0.0 to 3.5] | 1.0 [0.0 to 5.4]
  New or worsened joint pain: Grade 4 | 0 [0.0 to 3.4] | 0 [0.0 to 3.6] | 0 [0.0 to 3.3] | 0 [0.0 to 3.5] | 0 [0.0 to 3.6]

15. Primary Outcome: Cohort 2: Percentage of Participants With AEs From Study Vaccination Through 1 Month After Study Vaccination
Description: as for outcome 3
Time Frame: From study vaccination through 1 month after study vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2 (Group 1): 12-17 Years (BNT162b2 [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 2): 18-55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 3): 18-55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 60 mcg) | Cohort 2 (Group 4): >55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 5): >55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 60 mcg)
Number analyzed (Participants) | 107 | 103 | 110 | 106 | 102
Percentage of participants | 7.5 [3.3 to 14.2] | 2.9 [0.6 to 8.3] | 8.2 [3.8 to 15.0] | 3.8 [1.0 to 9.4] | 6.9 [2.8 to 13.6]

16. Primary Outcome: Cohort 2: Percentage of Participants With SAEs From Study Vaccination Through 6 Month After Study Vaccination
Description: An AE was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was an AE that resulted in death, was life-threatening, resulted in persistent disability/incapacity; constituted a congenital anomaly/birth defect; was important medical event; required inpatient hospitalization or prolongation of existing hospitalization.
Time Frame: From study vaccination through 6 months after study vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2 (Group 1): 12-17 Years (BNT162b2 [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 2): 18-55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 3): 18-55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 60 mcg) | Cohort 2 (Group 4): >55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 5): >55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 60 mcg)
Number analyzed (Participants) | 107 | 103 | 110 | 106 | 102
Percentage of participants | 0.9 [0.0 to 5.1] | 0 [0.0 to 3.5] | 0.9 [0.0 to 5.0] | 3.8 [1.0 to 9.4] | 0 [0.0 to 3.6]

17. Primary Outcome: Cohort 2 (Group 2 and 4) + Cohort 3 (Group 1 and Group 2): Percentage of Participants Reporting Local Reactions Within 7 Days After Study Vaccination
Description: Local reactions were recorded by participants in an e-diary. Local reactions included redness, swelling and pain at injection site. Redness and swelling were graded as mild: >2.0 to 5.0 cm, moderate: >5.0 to 10.0 cm, severe: >10.0 cm, grade 4 (potentially life threatening): necrosis or exfoliative dermatitis (redness) and necrosis (swelling). Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfered with daily activity, severe: prevented daily activity and grade 4 (potentially life threatening): emergency room visit or hospitalization for severe pain. Grade 4 reactions were classified by the investigator or medically qualified person. Local reactions reported as AEs in the case report form within 7 days after the study vaccination were also reported.
Time Frame: From Day 1 to Day 7 after study vaccination
Population: Safety population included all participants who received the study intervention and where appropriate informed consent was obtained. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and ''Number Analyzed'' signifies participants evaluable for the specified rows. The outcome measure was planned per protocol to be analyzed in participants combined from Cohort 2 (Group 2) + Cohort 3 (Group 1) and Cohort 2 (Group 4) + Cohort 3 (Group 2).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Cohort 2 (Group 2) + Cohort 3 (Group 1): 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg): Participants aged 18-55 years received BNT162b2 Bivalent (WT/OMI BA.4/BA.5) 30 mcg intramuscularly at Visit 1 (Day 1).
- Cohort 2 (Group 4) + Cohort 3 (Group 2): >55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg): Participants aged >55 years received BNT162b2 Bivalent (WT/OMI BA.4/BA.5) 30 mcg intramuscularly at Visit 1 (Day 1).
Arm/Group | Cohort 2 (Group 2) + Cohort 3 (Group 1): 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 4) + Cohort 3 (Group 2): >55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg)
Number analyzed (Participants) | 310 | 301
Percentage of participants
  Redness: Any: number analyzed (Participants) | 309 | 300
  Redness: Any | 6.5 [4.0 to 9.8] | 4.0 [2.1 to 6.9]
  Redness: Mild: number analyzed (Participants) | 309 | 300
  Redness: Mild | 4.9 [2.7 to 7.9] | 2.3 [0.9 to 4.7]
  Redness: Moderate: number analyzed (Participants) | 309 | 300
  Redness: Moderate | 1.6 [0.5 to 3.7] | 1.7 [0.5 to 3.8]
  Redness: Severe: number analyzed (Participants) | 309 | 300
  Redness: Severe | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Redness: Grade 4: number analyzed (Participants) | 309 | 300
  Redness: Grade 4 | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Swelling: Any: number analyzed (Participants) | 309 | 300
  Swelling: Any | 7.1 [4.5 to 10.6] | 2.7 [1.2 to 5.2]
  Swelling: Mild: number analyzed (Participants) | 309 | 300
  Swelling: Mild | 5.8 [3.5 to 9.1] | 1.7 [0.5 to 3.8]
  Swelling: Moderate: number analyzed (Participants) | 309 | 300
  Swelling: Moderate | 1.3 [0.4 to 3.3] | 1.0 [0.2 to 2.9]
  Swelling: Severe: number analyzed (Participants) | 309 | 300
  Swelling: Severe | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Swelling: Grade 4: number analyzed (Participants) | 309 | 300
  Swelling: Grade 4 | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Pain at the injection site: Any | 76.1 [71.0 to 80.8] | 57.1 [51.3 to 62.8]
  Pain at the injection site: Mild | 57.4 [51.7 to 63.0] | 48.8 [43.1 to 54.6]
  Pain at the injection site: Moderate | 18.7 [14.5 to 23.5] | 8.0 [5.2 to 11.6]
  Pain at the injection site: Severe | 0 [0.0 to 1.2] | 0.3 [0.0 to 1.8]
  Pain at the injection site: Grade 4 | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]

18. Primary Outcome: Cohort 2 (Group 2 and 4) + Cohort 3 (Group 1 and Group 2): Percentage of Participants Reporting Systemic Events Within 7 Days After Study Vaccination
Description: Systemic events were recorded by participants in an e-diary. Fever was oral temperature >= 38 deg C and categorized as >=38.0 to 38.4 deg C, >38.4 to 38.9 deg C, >38.9 to 40.0 deg C and >40.0 deg C. Fatigue, headache, chills, new or worsened muscle pain and new or worsened joint pain were graded as mild: did not interfere with activity, moderate: some interference with activity and severe: prevented daily routine activity. Vomiting was graded as mild: 1 to 2 times in 24 h, moderate: >2 times in 24h and severe: required intravenous hydration. Diarrhea was graded as mild: 2 to 3 loose stools in 24h, moderate: 4 to 5 loose stools in 24h and severe: 6 or more loose stools in 24h. For all systemic events except fever, Grade 4= emergency room visit or hospitalization. Grade 4 events were classified by the investigator/medically qualified person. Systemic events reported as AEs in the CRF within 7 days after vaccination were also reported.
Time Frame: From Day 1 to Day 7 after study vaccination
Population: Safety population included all participants who received the study intervention and where appropriate informed consent was obtained. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for the specified rows. The outcome measure was planned per protocol to be analyzed in participants combined from Cohort 2 (Group 2) + Cohort 3 (Group 1) and Cohort 2 (Group 4) + Cohort 3 (Group 2).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2 (Group 2) + Cohort 3 (Group 1): 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 4) + Cohort 3 (Group 2): >55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg)
Number analyzed (Participants) | 309 | 301
Percentage of participants
  Fever: Any: number analyzed (Participants) | 309 | 300
  Fever: Any | 4.9 [2.7 to 7.9] | 4.3 [2.3 to 7.3]
  Fever: >=38.0 deg C to 38.4 deg C: number analyzed (Participants) | 309 | 300
  Fever: >=38.0 deg C to 38.4 deg C | 2.9 [1.3 to 5.5] | 3.3 [1.6 to 6.0]
  Fever: >38.4 deg C to 38.9 deg C: number analyzed (Participants) | 309 | 300
  Fever: >38.4 deg C to 38.9 deg C | 1.9 [0.7 to 4.2] | 1.0 [0.2 to 2.9]
  Fever: >38.9 deg C to 40.0 deg C: number analyzed (Participants) | 309 | 300
  Fever: >38.9 deg C to 40.0 deg C | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Fever: >40.0 deg C: number analyzed (Participants) | 309 | 300
  Fever: >40.0 deg C | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Fatigue: Any | 61.2 [55.5 to 66.6] | 38.5 [33.0 to 44.3]
  Fatigue: Mild | 26.9 [22.0 to 32.2] | 18.6 [14.4 to 23.5]
  Fatigue: Moderate | 32.4 [27.2 to 37.9] | 18.6 [14.4 to 23.5]
  Fatigue: Severe | 1.9 [0.7 to 4.2] | 1.3 [0.4 to 3.4]
  Fatigue: Grade 4 | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Headache: Any: number analyzed (Participants) | 309 | 300
  Headache: Any | 46.6 [40.9 to 52.3] | 30.7 [25.5 to 36.2]
  Headache: Mild: number analyzed (Participants) | 309 | 300
  Headache: Mild | 28.2 [23.2 to 33.5] | 20.7 [16.2 to 25.7]
  Headache: Moderate: number analyzed (Participants) | 309 | 300
  Headache: Moderate | 17.8 [13.7 to 22.5] | 10.0 [6.8 to 14.0]
  Headache: Severe: number analyzed (Participants) | 309 | 300
  Headache: Severe | 0.6 [0.1 to 2.3] | 0 [0.0 to 1.2]
  Headache: Grade 4: number analyzed (Participants) | 309 | 300
  Headache: Grade 4 | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Chills: Any: number analyzed (Participants) | 309 | 300
  Chills: Any | 22.0 [17.5 to 27.0] | 12.0 [8.5 to 16.2]
  Chills: Mild: number analyzed (Participants) | 309 | 300
  Chills: Mild | 12.3 [8.9 to 16.5] | 7.0 [4.4 to 10.5]
  Chills: Moderate: number analyzed (Participants) | 309 | 300
  Chills: Moderate | 9.1 [6.1 to 12.8] | 4.7 [2.6 to 7.7]
  Chills: Severe: number analyzed (Participants) | 309 | 300
  Chills: Severe | 0.6 [0.1 to 2.3] | 0.3 [0.0 to 1.8]
  Chills: Grade 4: number analyzed (Participants) | 309 | 300
  Chills: Grade 4 | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Vomiting: Any: number analyzed (Participants) | 309 | 300
  Vomiting: Any | 1.9 [0.7 to 4.2] | 0.7 [0.1 to 2.4]
  Vomiting: Mild: number analyzed (Participants) | 309 | 300
  Vomiting: Mild | 1.6 [0.5 to 3.7] | 0.7 [0.1 to 2.4]
  Vomiting: Moderate: number analyzed (Participants) | 309 | 300
  Vomiting: Moderate | 0.3 [0.0 to 1.8] | 0 [0.0 to 1.2]
  Vomiting: Severe: number analyzed (Participants) | 309 | 300
  Vomiting: Severe | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Vomiting: Grade 4: number analyzed (Participants) | 309 | 300
  Vomiting: Grade 4 | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Diarrhea: Any | 10.7 [7.5 to 14.7] | 9.6 [6.5 to 13.5]
  Diarrhea: Mild | 8.7 [5.8 to 12.5] | 7.6 [4.9 to 11.2]
  Diarrhea: Moderate | 1.6 [0.5 to 3.7] | 2.0 [0.7 to 4.3]
  Diarrhea: Severe | 0.3 [0.0 to 1.8] | 0 [0.0 to 1.2]
  Diarrhea: Grade 4 | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  New or worsened muscle pain: Any: number analyzed (Participants) | 309 | 300
  New or worsened muscle pain: Any | 30.4 [25.3 to 35.9] | 18.0 [13.8 to 22.8]
  New or worsened muscle pain: Mild: number analyzed (Participants) | 309 | 300
  New or worsened muscle pain: Mild | 15.2 [11.4 to 19.7] | 10.0 [6.8 to 14.0]
  New or worsened muscle pain: Moderate: number analyzed (Participants) | 309 | 300
  New or worsened muscle pain: Moderate | 15.2 [11.4 to 19.7] | 8.0 [5.2 to 11.7]
  New or worsened muscle pain: Severe: number analyzed (Participants) | 309 | 300
  New or worsened muscle pain: Severe | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  New or worsened muscle pain: Grade 4: number analyzed (Participants) | 309 | 300
  New or worsened muscle pain: Grade 4 | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  New or worsened joint pain: Any: number analyzed (Participants) | 309 | 300
  New or worsened joint pain: Any | 14.9 [11.1 to 19.4] | 12.0 [8.5 to 16.2]
  New or worsened joint pain: Mild: number analyzed (Participants) | 309 | 300
  New or worsened joint pain: Mild | 6.8 [4.3 to 10.2] | 6.7 [4.1 to 10.1]
  New or worsened joint pain: Moderate: number analyzed (Participants) | 309 | 300
  New or worsened joint pain: Moderate | 8.1 [5.3 to 11.7] | 5.3 [3.1 to 8.5]
  New or worsened joint pain: Severe: number analyzed (Participants) | 309 | 300
  New or worsened joint pain: Severe | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  New or worsened joint pain: Grade 4: number analyzed (Participants) | 309 | 300
  New or worsened joint pain: Grade 4 | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]

19. Primary Outcome: Cohort 2 (Group 2 and 4) + Cohort 3 (Group 1 and Group 2): Percentage of Participants With AEs From Study Vaccination Through 1 Month After Study Vaccination
Description: as for outcome 3
Time Frame: From study vaccination through 1 month after study vaccination
Population: Safety population included all participants who received the study intervention and where appropriate informed consent was obtained. The outcome measure was planned per protocol to be analyzed in participants combined from Cohort 2 (Group 2) + Cohort 3 (Group 1) and Cohort 2 (Group 4) + Cohort 3 (Group 2).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2 (Group 2) + Cohort 3 (Group 1): 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 4) + Cohort 3 (Group 2): >55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg)
Number analyzed (Participants) | 313 | 306
Percentage of participants | 6.1 [3.7 to 9.3] | 6.9 [4.3 to 10.3]

20. Primary Outcome: Cohort 2 (Group 2 and 4) + Cohort 3 (Group 1 and Group 2): Percentage of Participants With SAEs From Study Vaccination Through 6 Month After Study Vaccination
Description: as for outcome 16
Time Frame: From study vaccination through 6 months after study vaccination
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2 (Group 2) + Cohort 3 (Group 1): 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 4) + Cohort 3 (Group 2): >55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg)
Number analyzed (Participants) | 313 | 306
Percentage of participants | 0.6 [0.1 to 2.3] | 3.3 [1.6 to 5.9]

21. Primary Outcome: GMR of Omicron (BA.4/BA.5)- NT of BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 30 mcg Cohort 2 (Group 4)/ Cohort 3 (Group 2) Combined in C4591044 Compared to NT of BNT162b2 30 mcg in C4591031 [NCT04955626]- 1 Month After Vaccination Among Participants >55 Years
Description: Model based GMT of OMI BA.4/BA.5 NTs induced by BNT162b2 Bivalent 30mcg groups of study C4591044 Cohort 2/3 combined and BNT162b2 30mcg of study C4591031 [NCT04955626] Substudy E among participants >55 years are reported as descriptive data. GMTs and 95% CIs were calculated by exponentiating least square (LS) means and corresponding CI based on analysis of logarithmically transformed NT using a linear regression model with terms of baseline NT (log scale) and vaccine group. Assay results below LLOQ were set to 0.5*LLOQ. Model based geometric mean ratio (GMR) are reported in statistical section: OMI BA.4/BA.5 NTs induced 1 month post BNT162b2 Bivalent vaccination in study C4591044 to 1 month post BNT162b2 vaccination in study C4591031 [NCT04955626] among participants >55 years. Outcome measure was planned per protocol to be analyzed in participants of Cohort 2 (Group 4) + Cohort 3 (Group 2) of C4591044 and BNT162b2 experienced participants of study C4591031 [NCT04955626] (control arm).
Time Frame: 1 month after study vaccination
Population: EIP: all assigned/ randomized participants who received study intervention to which they were randomized/assigned, had at least 1 valid, determinate immunogenicity result from blood sample collected within 28-42 days post vaccination and had no other important protocol deviations. Analysis was performed in participants with or without evidence of infection up to 1 month post vaccination. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- BNT162b2 30 mcg: C4591031 Substudy E: BNT162b2 experienced participants >55 years of age in study C4591031 [NCT04955626] received one dose (30 mcg) of BNT162b2 intramuscularly. As planned this group served as immunogenicity control arm and participants are not included in enrollment number of current C4591044 [NCT05472038] study.
Arm/Group | Cohort 2 (Group 4) + Cohort 3 (Group 2): >55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg) | BNT162b2 30 mcg: C4591031 Substudy E
Number analyzed (Participants) | 282 | 273
Titer | 3373.4 [3000.3 to 3793.0] | 1160.7 [1030.3 to 1307.7]
Statistical Analysis 1: Comparison: Cohort 2 (Group 4) + Cohort 3 (Group 2): >55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg) vs BNT162b2 30 mcg: C4591031 Substudy E; Test type: Superiority — Superiority based on GMR was declared if the lower limit of the 2-sided 95% CI for the GMR was greater than 1; Model-Based GMR = 2.91, 95% CI 2-sided [2.45 to 3.44]

22. Primary Outcome: Difference in Percentage of Participants With Seroresponse to OMI BA.4/BA.5 for BNT162b2 Bivalent[WT/OMI BA.4/BA.5]30mcg Cohort2(Group4)/Cohort3(Group2)Combined in C4591044 and BNT162b2 30mcg in C4591031-1 Month After Vaccination in Participants >55 Years
Description: Seroresponse: achieving >=4-fold rise in NTs from baseline (before study vaccination). If baseline measurement was below LLOQ, postvaccination measure of >= 4*LLOQ was considered seroresponse. Percentage of participants with seroresponse to OMI BA.4/BA.5 for BNT162b2 Bivalent 30 mcg in Study C4591044 [NCT05472038] Cohort 2/3 combined and BNT162b2 30 mcg in Study C4591031 [NCT04955626] Substudy E among participants >55 years of age are presented as descriptive data. Adjusted difference in seroresponse rate to OMI BA.4/BA.5 between BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg 1 month after vaccination in study C4591044 and 1 month after BNT162b2 vaccination in study C4591031 [NCT04955626] among participants >55 years of age is reported in statistical section. Outcome measure was planned per protocol to be analyzed in participants from Cohort 2 (Group 4) + Cohort 3 (Group 2) and control arm of BNT162b2 experienced participants >55 years of age from study C4591031 [NCT04955626] Substudy E.
Time Frame: 1 month after study vaccination
Population: EIP: all eligible, randomized participants who received study intervention to which they were randomized, had at least 1 valid and determinate immunogenicity result from blood sample collected within 28-42 days post study vaccination and had no other important protocol deviations. Analysis was performed in participants with or without evidence of infection up to 1 month post study vaccination. "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- BNT162b2 30 mcg: C4591031 Sub Study E: BNT162b2 experienced participants >55 years of age in study C4591031 [NCT04955626] received one dose (30 mcg) of BNT162b2 intramuscularly. As planned this group served as immunogenicity control arm and participants are not included in enrollment number of current C4591044 study.
Arm/Group | Cohort 2 (Group 4) + Cohort 3 (Group 2): >55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg) | BNT162b2 30 mcg: C4591031 Sub Study E
Number analyzed (Participants) | 282 | 273
Percentage of participants | 66.7 [60.8 to 72.1] | 46.5 [40.5 to 52.6]
Statistical Analysis 1: Comparison: Cohort 2 (Group 4) + Cohort 3 (Group 2): >55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg) vs BNT162b2 30 mcg: C4591031 Sub Study E; Test type: Non-Inferiority — Noninferiority based on seroresponse was declared if the lower limit of the 2-sided 95% CI for the difference in percentages of participants with seroresponse is >-5%; Adjusted Difference in Percentages = 26.77, 95% CI 2-sided [19.59 to 33.95] — Adjusted difference and 2-Sided CI based on the Miettinen and Nurminen method stratified by baseline NT category (< median,>= median) for difference in proportions. The median of baseline NT was calculated based on pooled data in 2 comparator groups

23. Primary Outcome: GMR of Omicron (BA.4/BA.5)- NTs of BNT162b2 Bivalent[WT/OMI BA.4/BA.5]30mcg Cohort2 (Group2)/Cohort3 (Group1)Combined for 18-55 Years Compared to BNT162b2 30mcg Cohort2 (Group4)/Cohort3 (Group2)Combined for >55 Years- 1 Month After Vaccination in C4591044
Description: Model based GMT of OMI BA.4/BA.5 NTs induced by BNT162b2 Bivalent 30 mcg groups of study C4591044 [NCT05472038] Cohort 2/3 combined in participants 18-55 years of age compared to participants >55 years of age are presented as descriptive data. GMTs and 2-sided 95% CIs were calculated by exponentiating LS means and corresponding CIs based on analysis of logarithmically transformed NT using a linear regression model with terms of baseline NT (log scale) and vaccine group. Assay results below LLOQ were set to 0.5*LLOQ. Model based GMR: OMI BA.4/BA.5 NTs induced 1 month after BNT162b2 Bivalent vaccination in study C4591044 among participants 18-55 years of age compared to participants >55 years of age is reported in statistical section. The outcome measure was planned per protocol to be analyzed in participants combined from Cohort 2 (Group 2) + Cohort 3 (Group 1) and Cohort 2 (Group 4) + Cohort 3 (Group 2).
Time Frame: 1 month after study vaccination
Population: EIP: all eligible, randomized participants who received study intervention to which they were randomized, had at least 1 valid and determinate immunogenicity result from blood sample collected within 28-42 days post study vaccination and had no other important protocol deviations. Analysis was performed in participants with or without prior evidence of infection up to 1 month post vaccination. "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- Cohort 2 (Group 2) + Cohort 3 (Group 1): 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg): Participants aged 18 to 55 years received BNT162b2 Bivalent (WT/OMI BA.4/BA.5) 30 mcg intramuscularly at Visit 1 (Day 1).
- Cohort 2 (Group 4) + Cohort 3 (Group 2): >55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg): Participants aged >55 years of age, received BNT162b2 Bivalent (WT/OMI BA.4/BA.5) 30 mcg intramuscularly at Visit 1 (Day 1).
Arm/Group | Cohort 2 (Group 2) + Cohort 3 (Group 1): 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 4) + Cohort 3 (Group 2): >55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg)
Number analyzed (Participants) | 294 | 282
Titer | 4254.2 [3779.6 to 4788.4] | 4344.4 [3850.2 to 4902.1]
Statistical Analysis 1: Comparison: Cohort 2 (Group 2) + Cohort 3 (Group 1): 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg) vs Cohort 2 (Group 4) + Cohort 3 (Group 2): >55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg); Test type: Non-Inferiority — Noninferiority based on the GMR was declared if the lower limit of the 2-sided 95% CI for the GMR is greater than 0.67 (1.5-fold criterion) and the point estimate of the GMR was >=0.8; Model-Based GMR = 0.98, 95% CI 2-sided [0.83 to 1.16] — GMR and 2-sided 95% CIs were calculated by exponentiating the difference of LS means and corresponding CIs based on the regression model included terms for baseline neutralizing titer and comparison group

24. Primary Outcome: Difference in Percentage of Participants With Seroresponse to OMI BA.4/BA.5 of BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg Cohort2 (Group2)/Cohort3 (Group1) 18-55 Years and Cohort2 (Group4)/Cohort3 (Group2) >55 Years- 1 Month After Vaccination in C4591044
Description: Seroresponse was defined as achieving >= 4-fold rise in NTs from baseline (before the study vaccination). If the baseline measurement was below the LLOQ, the postvaccination measure of >= 4*LLOQ was considered a seroresponse. Percentage of participants with seroresponse to OMI BA.4/BA.5 for BNT162b2 Bivalent 30 mcg in Study C4591044 [NCT05472038] Cohort 2/3 combined in participants 18-55 years of age compared to participants >55 years of age are presented as descriptive data. Adjusted difference in seroresponse rate to OMI BA.4/BA.5 between BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg 1 month after vaccination in study C4591044 in participants 18-55 years of age compared to participants >55 years of age is reported in statistical section. The outcome measure was planned per protocol to be analyzed in participants combined from Cohort 2 (Group 2) + Cohort 3 (Group 1) and Cohort 2 (Group 4) + Cohort 3 (Group 2).
Time Frame: 1 month after study vaccination
Population: EIP: all eligible, randomized participants who received study intervention to which they were randomized, had at least 1 valid and determinate immunogenicity result from blood sample collected within 28-42 days post study vaccination and had no important protocol deviations. Analysis was performed in participants with or without evidence of infection up to 1 month post study vaccination. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2 (Group 2) + Cohort 3 (Group 1): 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 4) + Cohort 3 (Group 2): >55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg)
Number analyzed (Participants) | 294 | 282
Percentage of participants | 61.2 [55.4 to 66.8] | 66.7 [60.8 to 72.1]
Statistical Analysis 1: Comparison: Cohort 2 (Group 2) + Cohort 3 (Group 1): 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg) vs Cohort 2 (Group 4) + Cohort 3 (Group 2): >55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg); Test type: Non-Inferiority — Noninferiority based on seroresponse was declared if the lower limit of the 2-sided 95% CI for the difference in percentages of participants with seroresponse is >-10%; Adjusted Difference in Percentages = -3.03, 95% CI 2-sided [-9.68 to 3.63] — 2-Sided CI based on Miettinen and Nurminen method stratified by baseline NT category(< median,>= median)for difference in percentage(seroresponse rate).Median of baseline neutralizing titers was calculated based on pooled data in 2 comparator groups

25. Primary Outcome: Cohort 2: GMT of SARS-CoV-2 Omicron Strain (BA.1 and BA.4/BA.5) and Reference Strain NTs at Baseline- Participants With or Without Evidence of Infection
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on student's t distribution). This outcome measure was planned per protocol to be analyzed in participants from Cohort 2 and control arms of BNT162b2 Bivalent (WT/OMI BA.1) experienced participants from study C4591031 [NCT04955626] Substudy E.
Time Frame: At baseline (before study vaccination)
Population: EIP: eligible, randomized participants received study intervention to which they were randomized, 1 valid, determinate immunogenicity result from blood sample collected within 28-42 days post study vaccination, no important protocol deviations. Analysis performed in participants with or without evidence of infection up to 1 month post study vaccination. Overall Number of Participants Analyzed= participants evaluable for outcome measure; Number Analyzed= participants evaluable for specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- Cohort 2 (Group 1): 12-17 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg): Participants aged 12-17 years received BNT162b2 Bivalent (WT/OMI BA.4/BA.5) 30 mcg intramuscularly at Visit 1 (Day 1).
- Cohort 2 (Group 2): 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg): Participants aged 18-55 years received BNT162b2 Bivalent (WT/OMI BA.4/BA.5) 30 mcg intramuscularly at Visit 1 (Day 1).
- Cohort 2 (Group 3): 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 60 mcg): Participants aged 18-55 years received BNT162b2 Bivalent (WT/OMI BA.4/BA.5) 60 mcg intramuscularly at Visit 1 (Day 1).
- Cohort 2 (Group 4): >55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg): Participants aged >55 years received BNT162b2 Bivalent (WT/OMI BA.4/BA.5) 30 mcg intramuscularly at Visit 1 (Day 1).
- Cohort 2 (Group 5): >55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 60 mcg): Participants aged >55 years received BNT162b2 Bivalent (WT/OMI BA.4/BA.5) 60 mcg intramuscularly at Visit 1 (Day 1).
- 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.1] 30 mcg): C4591031 Substudy E: BNT162b2 experienced participants 18-55 years of age in study C4591031 [NCT04955626] received one dose (30 mcg) of BNT162b2 intramuscularly. As planned this group served as immunogenicity control arm and participants are not included in enrollment number of current C4591044 [NCT05472038] study.
- 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.1] 60 mcg): C4591031 Substudy E: BNT162b2 experienced participants 18-55 years of age in study C4591031 [NCT04955626] received one dose (60 mcg) of BNT162b2 intramuscularly. As planned this group served as immunogenicity control arm and participants are not included in enrollment number of current C4591044 [NCT05472038] study.
- >55 Years (BNT162b2 Bivalent [WT/OMI BA.1] 30 mcg): C4591031 Substudy E: BNT162b2 experienced participants >55 years of age in study C4591031 [NCT04955626] received one dose (30 mcg) of BNT162b2 intramuscularly. As planned this group served as immunogenicity control arm and participants are not included in enrollment number of current C4591044 [NCT05472038] study.
- >55 Years (BNT162b2 Bivalent [WT/OMI BA.1] 60 mcg): C4591031 Substudy E: BNT162b2 experienced participants >55 years of age in study C4591031 [NCT04955626] received one dose (60 mcg) of BNT162b2 intramuscularly. As planned this group served as immunogenicity control arm and participants are not included in enrollment number of current C4591044 [NCT05472038] study.
Arm/Group | Cohort 2 (Group 1): 12-17 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 2): 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 3): 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 60 mcg) | Cohort 2 (Group 4): >55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 5): >55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 60 mcg) | 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.1] 30 mcg): C4591031 Substudy E | 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.1] 60 mcg): C4591031 Substudy E | >55 Years (BNT162b2 Bivalent [WT/OMI BA.1] 30 mcg): C4591031 Substudy E | >55 Years (BNT162b2 Bivalent [WT/OMI BA.1] 60 mcg): C4591031 Substudy E
Number analyzed (Participants) | 105 | 95 | 102 | 102 | 98 | 100 | 100 | 100 | 100
Titer
  Omicron BA.4/BA.5: number analyzed (Participants) | 104 | 95 | 102 | 101 | 98 | 100 | 100 | 99 | 100
  Omicron BA.4/BA.5 | 1105.8 [835.1 to 1464.3] | 338.3 [238.1 to 480.7] | 607.0 [433.2 to 850.6] | 301.9 [215.6 to 422.8] | 582.4 [397.6 to 853.1] | 151.5 [113.4 to 202.3] | 420.6 [312.7 to 565.6] | 225.4 [164.1 to 309.6] | 249.6 [180.5 to 345.2]
  Omicron BA.1: number analyzed (Participants) | 105 | 95 | 102 | 102 | 96 | 100 | 98 | 100 | 97
  Omicron BA.1 | 1190.5 [921.8 to 1537.5] | 346.0 [240.0 to 498.9] | 653.1 [466.3 to 914.8] | 365.1 [260.8 to 511.1] | 581.2 [392.5 to 860.6] | 194.6 [142.4 to 266.0] | 492.4 [351.5 to 689.9] | 316.3 [215.9 to 463.4] | 285.6 [195.8 to 416.5]
  Reference-strain: number analyzed (Participants) | 105 | 95 | 101 | 101 | 98 | 100 | 100 | 100 | 100
  Reference-strain | 6863.3 [5587.8 to 8430.1] | 2349.0 [1693.4 to 3258.4] | 4287.4 [3245.6 to 5663.8] | 2643.1 [1990.8 to 3509.1] | 4324.8 [3099.0 to 6035.4] | 1338.4 [1056.9 to 1695.1] | 3933.2 [3058.0 to 5058.9] | 1985.7 [1510.1 to 2611.0] | 2509.3 [1906.8 to 3302.3]

26. Primary Outcome: Cohort 2: GMT of SARS-CoV-2 Omicron Strain (BA.1 and BA.4/BA.5) and Reference Strain NTs at 1 Month- Participants With or Without Evidence of Infection
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on student's t distribution). This outcome measure was planned per protocol to be analyzed in participants from Cohort 2 and control arms of BNT162b2 experienced participants from study C4591031 [NCT04955626] Substudy E.
Time Frame: 1 month after the study vaccination
Population: EIP: eligible, randomized participants received study intervention to which they were randomized, 1 valid, determinate immunogenicity result from blood sample collected within 28-42 days post study vaccination, no important protocol deviations. Analysis performed in participants with or without evidence of infection up to 1 month post study vaccination. Here, ''Number Analyzed'' signifies participants evaluable for specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- 18-55 Years (BNT162b2 30 mcg): C4591031 Substudy E: BNT162b2 experienced participants 18-55 years of age in study C4591031 [NCT04955626] received one dose (30 mcg) of BNT162b2 intramuscularly. As planned this group served as immunogenicity control arm and participants are not included in enrollment number of current C4591044 [NCT05472038] study.
- 18-55 Years (BNT162b2 60 mcg): C4591031 Substudy E: BNT162b2 experienced participants 18-55 years of age in study C4591031 [NCT04955626] received one dose (60 mcg) of BNT162b2 intramuscularly. As planned this group served as immunogenicity control arm and participants are not included in enrollment number of current C4591044 [NCT05472038] study.
- >55 Years (BNT162b2 30 mcg): C4591031 Substudy E: BNT162b2 experienced participants >55 years of age in study C4591031 [NCT04955626] received one dose (30 mcg) of BNT162b2 intramuscularly. As planned this group served as immunogenicity control arm and participants are not included in enrollment number of current C4591044 [NCT05472038] study.
- >55 Years (BNT162b2 60 mcg): C4591031 Substudy E: BNT162b2 experienced participants >55 years of age in study C4591031 [NCT04955626] received one dose (60 mcg) of BNT162b2 intramuscularly. As planned this group served as immunogenicity control arm and participants are not included in enrollment number of current C4591044 [NCT05472038] study.
Arm/Group | Cohort 2 (Group 1): 12-17 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 2): 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 3): 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 60 mcg) | Cohort 2 (Group 4): >55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 5): >55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 60 mcg) | 18-55 Years (BNT162b2 30 mcg): C4591031 Substudy E | 18-55 Years (BNT162b2 60 mcg): C4591031 Substudy E | >55 Years (BNT162b2 30 mcg): C4591031 Substudy E | >55 Years (BNT162b2 60 mcg): C4591031 Substudy E
Number analyzed (Participants) | 105 | 95 | 102 | 102 | 99 | 100 | 100 | 100 | 100
Titer
  Omicron BA.4/BA.5 | 8212.8 [6807.3 to 9908.7] | 2839.0 [2150.0 to 3748.8] | 5454.2 [4292.2 to 6930.8] | 3019.8 [2327.5 to 3918.0] | 5472.8 [3930.9 to 7619.6] | 1072.0 [816.1 to 1408.1] | 2525.2 [1970.5 to 3236.0] | 943.4 [733.4 to 1213.6] | 1520.9 [1196.0 to 1934.0]
  Omicron BA.1: number analyzed (Participants) | 105 | 95 | 101 | 102 | 99 | 100 | 99 | 100 | 100
  Omicron BA.1 | 6687.6 [5617.0 to 7962.3] | 2407.2 [1884.9 to 3074.2] | 4112.4 [3263.6 to 5181.9] | 2656.1 [2089.6 to 3376.3] | 4264.0 [3247.9 to 5597.9] | 1819.0 [1401.6 to 2360.6] | 3143.8 [2486.9 to 3974.1] | 1617.7 [1274.7 to 2053.0] | 1936.9 [1489.4 to 2518.8]
  Reference-strain: number analyzed (Participants) | 105 | 95 | 102 | 102 | 99 | 99 | 100 | 100 | 99
  Reference-strain | 23641.3 [20473.1 to 27299.8] | 11919.3 [9839.1 to 14439.3] | 18614.7 [15754.1 to 21994.7] | 12103.8 [9992.0 to 14662.0] | 22982.3 [18524.3 to 28513.3] | 6913.9 [5690.4 to 8400.5] | 14685.8 [12301.1 to 17532.8] | 7128.6 [5954.4 to 8534.3] | 11106.5 [8956.8 to 13772.2]

27. Primary Outcome: Cohort 2: GMFR of SARS-CoV-2 Omicron Strain (BA.1 and BA.4/BA.5) and Reference Strain- NTs From Before the Study Vaccination to 1 Month After the Study Vaccination- Participants With or Without Evidence of Infection
Description: GMFR from before the study vaccination to 1 month after the study vaccination for each strain-specific neutralizing titer was reported in this outcome measure. GMFRs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the student-t distribution). Assay results below the LLOQ were set to 0.5*LLOQ in the analysis. This outcome measure was planned per protocol to be analyzed in participants from Cohort 2 and control arms of BNT162b2 experienced participants from study C4591031 [NCT04955626] Substudy E.
Time Frame: From before the study vaccination to 1 month after the study vaccination
Population: as for outcome 25
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Cohort 2 (Group 1): 12-17 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 2): 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 3): 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 60 mcg) | Cohort 2 (Group 4): >55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 5): >55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 60 mcg) | 18-55 Years (BNT162b2 30 mcg): C4591031 Substudy E | 18-55 Years (BNT162b2 60 mcg): C4591031 Substudy E | >55 Years (BNT162b2 30 mcg): C4591031 Substudy E | >55 Years (BNT162b2 60 mcg): C4591031 Substudy E
Number analyzed (Participants) | 105 | 95 | 102 | 102 | 98 | 100 | 100 | 100 | 100
Fold rise
  Omicron BA.4/BA.5: number analyzed (Participants) | 104 | 95 | 102 | 101 | 98 | 100 | 100 | 99 | 100
  Omicron BA.4/BA.5 | 7.6 [6.0 to 9.6] | 8.4 [6.3 to 11.1] | 9.0 [6.9 to 11.8] | 10.0 [7.5 to 13.3] | 9.3 [6.8 to 12.8] | 7.1 [5.7 to 8.9] | 6.0 [4.7 to 7.7] | 4.2 [3.4 to 5.2] | 6.1 [4.7 to 7.9]
  Omicron BA.1: number analyzed (Participants) | 105 | 95 | 101 | 102 | 96 | 100 | 97 | 100 | 97
  Omicron BA.1 | 5.6 [4.6 to 6.9] | 7.0 [5.3 to 9.1] | 6.3 [4.9 to 8.2] | 7.3 [5.6 to 9.5] | 7.3 [5.4 to 9.7] | 9.3 [7.3 to 12.0] | 6.4 [4.9 to 8.3] | 5.1 [3.9 to 6.6] | 6.8 [5.1 to 9.1]
  Reference-strain: number analyzed (Participants) | 105 | 95 | 101 | 101 | 98 | 99 | 100 | 100 | 99
  Reference-strain | 3.4 [2.9 to 4.1] | 5.1 [3.9 to 6.6] | 4.3 [3.4 to 5.5] | 4.6 [3.7 to 5.8] | 5.4 [4.0 to 7.1] | 5.2 [4.3 to 6.3] | 3.7 [3.0 to 4.6] | 3.6 [2.9 to 4.4] | 4.4 [3.5 to 5.6]

28. Primary Outcome: Cohort 2: Percentage of Participants With Seroresponse to SARS-CoV-2 Omicron Strain (BA.1 and BA.4/BA.5) and Reference Strain- NTs at 1 Month After Study Vaccination- Participants With or Without Evidence of Infection
Description: Seroresponse was defined as achieving >= 4-fold rise in NTs from baseline (before the study vaccination). If the baseline measurement was below the LLOQ, the postvaccination measure of >= 4*LLOQ was considered a seroresponse. Percentage of participants with seroresponse to OMI BA.4/BA.5 for BNT162b2 Bivalent 30 and 60 mcg in Study C4591044 [NCT05472038] Cohort 2 and BNT162b2 30 mcg in Study C4591031 [NCT04955626] Substudy E are presented as descriptive data. This outcome measure was planned per protocol to be analyzed in participants from Cohort 2 and control arms of BNT162b2 experienced participants 18-55 years of age and >55 years of age from study C4591031 [NCT04955626] Substudy E.
Time Frame: 1 month after the study vaccination
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2 (Group 1): 12-17 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 2): 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 3): 18-55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 60 mcg) | Cohort 2 (Group 4): >55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 5): >55 Years (BNT162b2 Bivalent [WT/OMI BA.4/BA.5] 60 mcg) | 18-55 Years (BNT162b2 30 mcg): C4591031 Substudy E | 18-55 Years (BNT162b2 60 mcg): C4591031 Substudy E | >55 Years (BNT162b2 30 mcg): C4591031 Substudy E | >55 Years (BNT162b2 60 mcg): C4591031 Substudy E
Number analyzed (Participants) | 105 | 95 | 102 | 102 | 98 | 100 | 100 | 100 | 100
Percentage of participants
  Omicron BA.4/BA.5: number analyzed (Participants) | 104 | 95 | 102 | 101 | 98 | 100 | 100 | 99 | 100
  Omicron BA.4/BA.5 | 66.3 [56.4 to 75.3] | 64.2 [53.7 to 73.8] | 66.7 [56.6 to 75.7] | 71.3 [61.4 to 79.9] | 63.3 [52.9 to 72.8] | 62.0 [51.7 to 71.5] | 59.0 [48.7 to 68.7] | 37.4 [27.9 to 47.7] | 53.0 [42.8 to 63.1]
  Omicron BA.1: number analyzed (Participants) | 105 | 95 | 101 | 102 | 96 | 100 | 97 | 100 | 97
  Omicron BA.1 | 63.8 [53.9 to 73.0] | 54.7 [44.2 to 65.0] | 60.4 [50.2 to 70.0] | 63.7 [53.6 to 73.0] | 65.6 [55.2 to 75.0] | 75.0 [65.3 to 83.1] | 56.7 [46.3 to 66.7] | 52.0 [41.8 to 62.1] | 58.8 [48.3 to 68.7]
  Reference-strain: number analyzed (Participants) | 105 | 95 | 101 | 101 | 98 | 99 | 100 | 100 | 99
  Reference-strain | 41.0 [31.5 to 51.0] | 49.5 [39.1 to 59.9] | 51.5 [41.3 to 61.6] | 50.5 [40.4 to 60.6] | 55.1 [44.7 to 65.2] | 59.6 [49.3 to 69.3] | 41.0 [31.3 to 51.3] | 41.0 [31.3 to 51.3] | 44.4 [34.5 to 54.8]

29. Secondary Outcome: GMR of the Reference-Strain- NTs of BNT162b2 [WT/OMI BA.4/BA.5] 30mcg Cohort 2 (Group 4)/ Cohort 3 (Group 2) Combined in C4591044 Compared to NT of BNT162b2 30mcg in C4591031 [NCT04955626] >55 Years of Age- 1 Month After Vaccination
Description: Model based GMT of reference strain NTs induced by BNT162b2 Bivalent 30mcg groups of study C4591044 [NCT05472038] Cohort 2/3 combined and BNT162b2 30 mcg of study C4591031 [NCT04955626] Substudy E among participants >55 years of age presented as descriptive data. GMTs, 2-sided 95% CIs calculated by exponentiating LS means, corresponding CIs based on analysis of logarithmically transformed NT using linear regression model with terms of baseline NT (log scale), vaccine group. Assay results below LLOQ set to 0.5*LLOQ. Model based GMR: OMI BA.4/BA.5 NTs induced 1 month after BNT162b2 Bivalent vaccination in study C4591044 to 1 month after BNT162b2 vaccination in study C4591031 [NCT04955626] among participants >55 years of age reported in statistical section. Outcome measure was planned per protocol to be analyzed in participants from Cohort 2 (Group 4) + Cohort 3 (Group 2) and control arm of BNT162b2 experienced participants >55 years of age from study C4591031 [NCT04955626] Substudy E.
Time Frame: 1 month after study vaccination
Population: EIP included all assigned/ randomized participants who received study intervention to which they were randomized/assigned, had at least 1 valid and determinate immunogenicity result from blood sample collected within 28-42 days post the vaccination and had no other important protocol deviations. Analysis in participants with or without prior evidence of infection up to 1 month post vaccination. "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- Cohort 2 (Group 4) + Cohort 3 (Group 2): >55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 30 mcg): Participants aged >55 years received BNT162b2 Bivalent (WT/OMI BA.4/BA.5) 30 mcg intramuscularly at Visit 1 (Day 1).
Arm/Group | Cohort 2 (Group 4) + Cohort 3 (Group 2): >55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 30 mcg) | BNT162b2 30 mcg: C4591031 Substudy E
Number analyzed (Participants) | 284 | 287
Titer | 15361.6 [14082.9 to 16756.5] | 11117.2 [10196.4 to 12121.1]
Statistical Analysis 1: Comparison: Cohort 2 (Group 4) + Cohort 3 (Group 2): >55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 30 mcg) vs BNT162b2 30 mcg: C4591031 Substudy E; Test type: Non-Inferiority — [test comment as in outcome 23, analysis 1]; Model-Based GMR = 1.38, 95% CI 2-sided [1.22 to 1.56] — [estimate comment as in outcome 23, analysis 1]

30. Secondary Outcome: Cohort 2 (Group 2) + Cohort 3 (Group 1) Combined and Cohort 2 (Group 4) + Cohort 3 (Group 2) Combined: GMT of Omicron BA.4/BA.5 and Reference Strain NT at Baseline and 1 Month After the Study Vaccination
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on student's t distribution). This outcome measure was planned per protocol to be analyzed in participants from Cohort 2 (Group 2) + Cohort 3 (Group 1), Cohort 2 (Group 4) + Cohort 3 (Group 2) and control arm of BNT162b2 experienced participants >55 years of age from study C4591031 [NCT04955626] Substudy E.
Time Frame: At baseline and 1 month after study vaccination
Population: EIP included all assigned/ randomized participants who received study intervention to which they were randomized/assigned, had at least 1 valid and determinate immunogenicity result from blood sample collected within 28-42 days post the vaccination and had no other important protocol deviations. Analysis was performed in participants with or without evidence of infection up to 1 month post study vaccination. Here, ''Number Analyzed'' signifies participants evaluable for specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- Cohort 2 (Group 2) + Cohort 3 (Group 1): 18-55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 30 mcg): Participants aged 18-55 years received BNT162b2 Bivalent (WT/OMI BA.4/BA.5) 30 mcg intramuscularly at Visit 1 (Day 1).
Arm/Group | Cohort 2 (Group 2) + Cohort 3 (Group 1): 18-55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 4) + Cohort 3 (Group 2): >55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 30 mcg) | BNT162b2 30 mcg: C4591031 Substudy E
Number analyzed (Participants) | 297 | 286 | 289
Titer
  Omicron BA.4/BA.5 at baseline: number analyzed (Participants) | 294 | 284 | 278
  Omicron BA.4/BA.5 at baseline | 569.6 [471.4 to 688.2] | 458.2 [365.2 to 574.8] | 205.4 [170.3 to 247.7]
  Omicron BA.4/BA.5 at 1 Month: number analyzed (Participants) | 297 | 284 | 282
  Omicron BA.4/BA.5 at 1 Month | 4455.9 [3851.7 to 5154.8] | 4158.1 [3554.8 to 4863.8] | 938.9 [802.3 to 1098.8]
  Reference strain at baseline: number analyzed (Participants) | 296 | 284 | 287
  Reference strain at baseline | 4017.3 [3430.7 to 4704.1] | 3690.6 [3082.2 to 4419.0] | 2699.9 [2291.7 to 3180.9]
  Reference strain at 1 Month: number analyzed (Participants) | 296 | 286 | 289
  Reference strain at 1 Month | 16323.3 [14686.5 to 18142.6] | 16250.1 [14499.2 to 18212.4] | 10415.5 [9366.7 to 11581.8]

31. Secondary Outcome: Cohort 2 (Group 2) + Cohort 3 (Group 1) Combined and Cohort 2 (Group 4) + Cohort 3 (Group 2) Combined: GMFR of SARS-CoV-2 Omicron Strain (BA.4/BA.5) and Reference Strain- NTs From Before the Study Vaccination to 1 Month After the Study Vaccination
Description: GMFRs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ in the analysis. GMFR from before the study vaccination to 1 month after study vaccination for Omicron BA.4/BA.5 and reference strain neutralizing titer was reported in this outcome measure. This outcome measure was planned per protocol to be analyzed in participants from Cohort 2 (Group 2) + Cohort 3 (Group 1), Cohort 2 (Group 4) + Cohort 3 (Group 2) and control arm of BNT162b2 experienced participants >55 years of age from study C4591031 [NCT04955626] Substudy E.
Time Frame: From before the study vaccination to 1 month after study vaccination
Population: as for outcome 30
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Cohort 2 (Group 2) + Cohort 3 (Group 1): 18-55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 4) + Cohort 3 (Group 2): >55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 30 mcg) | BNT162b2 30 mcg: C4591031 Substudy E
Number analyzed (Participants) | 295 | 284 | 287
Fold rise
  Omicron BA.4/BA.5: number analyzed (Participants) | 294 | 282 | 273
  Omicron BA.4/BA.5 | 7.8 [6.7 to 9.2] | 8.9 [7.5 to 10.6] | 4.6 [4.0 to 5.2]
  Reference strain | 4.1 [3.6 to 4.6] | 4.4 [3.8 to 5.1] | 3.9 [3.4 to 4.4]

32. Secondary Outcome: Cohort 2 (Group 2) + Cohort 3 (Group 1) Combined and Cohort 2 (Group 4) + Cohort 3 (Group 2) Combined: Percentages of Participants With Seroresponse to SARS-CoV-2 Omicron Strain (BA.4/BA.5) and Reference Strain- NTs at 1 Month After the Study Vaccination
Description: Seroresponse was defined as achieving >= 4-fold rise in NTs from baseline (before the study vaccination). If the baseline measurement was below the LLOQ, the postvaccination measure of >= 4*LLOQ was considered a seroresponse. Percentage of participants with seroresponse to OMI BA.4/BA.5 for BNT162b2 Bivalent 30 mcg in Study C4591044 [NCT05472038] Cohort 2/3 combined and BNT162b2 30 mcg in Study C4591031 [NCT04955626] Substudy E among participants >55 years of age are presented as descriptive data. This outcome measure was planned per protocol to be analyzed in participants from Cohort 2 (Group 2) + Cohort 3 (Group 1), Cohort 2 (Group 4) + Cohort 3 (Group 2) and control arm of BNT162b2 experienced participants >55 years of age from study C4591031 [NCT04955626] Substudy E.
Time Frame: 1 month after the study vaccination
Population: EIP was analyzed. Analysis was performed in EIP with or without evidence of infection up to 1 month post study vaccination. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and ''Number Analyzed'' signifies participants evaluable for specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2 (Group 2) + Cohort 3 (Group 1): 18-55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 30 mcg) | Cohort 2 (Group 4) + Cohort 3 (Group 2): >55 Years (BNT162b2 [WT/OMI BA.4/BA.5] 30 mcg) | BNT162b2 30 mcg: C4591031 Substudy E
Number analyzed (Participants) | 295 | 284 | 287
Percentage of participants
  Omicron BA.4/BA.5: number analyzed (Participants) | 294 | 282 | 273
  Omicron BA.4/BA.5 | 61.2 [55.4 to 66.8] | 66.7 [60.8 to 72.1] | 46.5 [40.5 to 52.6]
  Reference strain | 44.1 [38.3 to 49.9] | 45.8 [39.9 to 51.8] | 48.1 [42.2 to 54.0]

33. Primary Outcome: Cohort 4: Percentage of Participants Reporting Local Reactions Within 7 Days After Study Vaccination
Description: as for outcome 17
Time Frame: From Day 1 to Day 7 after study vaccination
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 4: 18-55 Years (BNT162b2 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b5 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b6 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b7 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b7 Monovalent [OMI BA.4/ BA.5] 30 mcg)
Number analyzed (Participants) | 62 | 61 | 60 | 60 | 63
Percentage of participants
  Redness: Any | 4.8 [1.0 to 13.5] | 3.3 [0.4 to 11.3] | 5.0 [1.0 to 13.9] | 1.7 [0.0 to 8.9] | 1.6 [0.0 to 8.5]
  Redness: Mild | 3.2 [0.4 to 11.2] | 3.3 [0.4 to 11.3] | 5.0 [1.0 to 13.9] | 1.7 [0.0 to 8.9] | 1.6 [0.0 to 8.5]
  Redness: Moderate | 1.6 [0.0 to 8.7] | 0 [0.0 to 5.9] | 0 [0.0 to 6.0] | 0 [0.0 to 6.0] | 0 [0.0 to 5.7]
  Redness: Severe | 0 [0.0 to 5.8] | 0 [0.0 to 5.9] | 0 [0.0 to 6.0] | 0 [0.0 to 6.0] | 0 [0.0 to 5.7]
  Redness: Grade 4 | 0 [0.0 to 5.8] | 0 [0.0 to 5.9] | 0 [0.0 to 6.0] | 0 [0.0 to 6.0] | 0 [0.0 to 5.7]
  Swelling: Any | 1.6 [0.0 to 8.7] | 3.3 [0.4 to 11.3] | 6.7 [1.8 to 16.2] | 3.3 [0.4 to 11.5] | 3.2 [0.4 to 11.0]
  Swelling: Mild | 0 [0.0 to 5.8] | 0 [0.0 to 5.9] | 6.7 [1.8 to 16.2] | 3.3 [0.4 to 11.5] | 3.2 [0.4 to 11.0]
  Swelling: Moderate | 1.6 [0.0 to 8.7] | 3.3 [0.4 to 11.3] | 0 [0.0 to 6.0] | 0 [0.0 to 6.0] | 0 [0.0 to 5.7]
  Swelling: Severe | 0 [0.0 to 5.8] | 0 [0.0 to 5.9] | 0 [0.0 to 6.0] | 0 [0.0 to 6.0] | 0 [0.0 to 5.7]
  Swelling: Grade 4 | 0 [0.0 to 5.8] | 0 [0.0 to 5.9] | 0 [0.0 to 6.0] | 0 [0.0 to 6.0] | 0 [0.0 to 5.7]
  Pain at injection site: Any | 85.5 [74.2 to 93.1] | 88.5 [77.8 to 95.3] | 76.7 [64.0 to 86.6] | 76.7 [64.0 to 86.6] | 84.1 [72.7 to 92.1]
  Pain at injection site: Mild | 64.5 [51.3 to 76.3] | 65.6 [52.3 to 77.3] | 68.3 [55.0 to 79.7] | 61.7 [48.2 to 73.9] | 68.3 [55.3 to 79.4]
  Pain at injection site: Moderate | 21.0 [11.7 to 33.2] | 21.3 [11.9 to 33.7] | 8.3 [2.8 to 18.4] | 15.0 [7.1 to 26.6] | 15.9 [7.9 to 27.3]
  Pain at injection site: Severe | 0 [0.0 to 5.8] | 1.6 [0.0 to 8.8] | 0 [0.0 to 6.0] | 0 [0.0 to 6.0] | 0 [0.0 to 5.7]
  Pain at injection site: Grade 4 | 0 [0.0 to 5.8] | 0 [0.0 to 5.9] | 0 [0.0 to 6.0] | 0 [0.0 to 6.0] | 0 [0.0 to 5.7]

34. Primary Outcome: Cohort 4: Percentage of Participants Reporting Systemic Events Within 7 Days After Study Vaccination
Description: as for outcome 14
Time Frame: From Day 1 to Day 7 after study vaccination
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 4: 18-55 Years (BNT162b2 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b5 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b6 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b7 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b7 Monovalent [OMI BA.4/ BA.5] 30 mcg)
Number analyzed (Participants) | 62 | 61 | 60 | 60 | 63
Percentage of participants
  Fever: Any | 6.5 [1.8 to 15.7] | 6.6 [1.8 to 15.9] | 10.0 [3.8 to 20.5] | 5.0 [1.0 to 13.9] | 9.5 [3.6 to 19.6]
  Fever: >=38.0 deg C to 38.4 deg C | 3.2 [0.4 to 11.2] | 6.6 [1.8 to 15.9] | 5.0 [1.0 to 13.9] | 5.0 [1.0 to 13.9] | 4.8 [1.0 to 13.3]
  Fever: >38.4 deg C to 38.9 deg C | 3.2 [0.4 to 11.2] | 0 [0.0 to 5.9] | 3.3 [0.4 to 11.5] | 0 [0.0 to 6.0] | 1.6 [0.0 to 8.5]
  Fever: >38.9 deg C to 40.0 deg C | 0 [0.0 to 5.8] | 0 [0.0 to 5.9] | 1.7 [0.0 to 8.9] | 0 [0.0 to 6.0] | 3.2 [0.4 to 11.0]
  Fever: >40.0 deg C | 0 [0.0 to 5.8] | 0 [0.0 to 5.9] | 0 [0.0 to 6.0] | 0 [0.0 to 6.0] | 0 [0.0 to 5.7]
  Fatigue: Any | 61.3 [48.1 to 73.4] | 63.9 [50.6 to 75.8] | 73.3 [60.3 to 83.9] | 66.7 [53.3 to 78.3] | 54.0 [40.9 to 66.6]
  Fatigue: Mild | 25.8 [15.5 to 38.5] | 29.5 [18.5 to 42.6] | 38.3 [26.1 to 51.8] | 35.0 [23.1 to 48.4] | 17.5 [9.1 to 29.1]
  Fatigue: Moderate | 35.5 [23.7 to 48.7] | 34.4 [22.7 to 47.7] | 33.3 [21.7 to 46.7] | 30.0 [18.8 to 43.2] | 34.9 [23.3 to 48.0]
  Fatigue: Severe | 0 [0.0 to 5.8] | 0 [0.0 to 5.9] | 1.7 [0.0 to 8.9] | 1.7 [0.0 to 8.9] | 1.6 [0.0 to 8.5]
  Fatigue: Grade 4 | 0 [0.0 to 5.8] | 0 [0.0 to 5.9] | 0 [0.0 to 6.0] | 0 [0.0 to 6.0] | 0 [0.0 to 5.7]
  Headache: Any | 59.7 [46.4 to 71.9] | 36.1 [24.2 to 49.4] | 41.7 [29.1 to 55.1] | 46.7 [33.7 to 60.0] | 39.7 [27.6 to 52.8]
  Headache: Mild | 38.7 [26.6 to 51.9] | 16.4 [8.2 to 28.1] | 23.3 [13.4 to 36.0] | 23.3 [13.4 to 36.0] | 22.2 [12.7 to 34.5]
  Headache: Moderate | 17.7 [9.2 to 29.5] | 19.7 [10.6 to 31.8] | 18.3 [9.5 to 30.4] | 21.7 [12.1 to 34.2] | 17.5 [9.1 to 29.1]
  Headache: Severe | 3.2 [0.4 to 11.2] | 0 [0.0 to 5.9] | 0 [0.0 to 6.0] | 1.7 [0.0 to 8.9] | 0 [0.0 to 5.7]
  Headache: Grade 4 | 0 [0.0 to 5.8] | 0 [0.0 to 5.9] | 0 [0.0 to 6.0] | 0 [0.0 to 6.0] | 0 [0.0 to 5.7]
  Chills: Any | 22.6 [12.9 to 35.0] | 18.0 [9.4 to 30.0] | 28.3 [17.5 to 41.4] | 13.3 [5.9 to 24.6] | 19.0 [10.2 to 30.9]
  Chills: Mild | 11.3 [4.7 to 21.9] | 11.5 [4.7 to 22.2] | 18.3 [9.5 to 30.4] | 8.3 [2.8 to 18.4] | 12.7 [5.6 to 23.5]
  Chills: Moderate | 11.3 [4.7 to 21.9] | 6.6 [1.8 to 15.9] | 10.0 [3.8 to 20.5] | 5.0 [1.0 to 13.9] | 6.3 [1.8 to 15.5]
  Chills: Severe | 0 [0.0 to 5.8] | 0 [0.0 to 5.9] | 0 [0.0 to 6.0] | 0 [0.0 to 6.0] | 0 [0.0 to 5.7]
  Chills: Grade 4 | 0 [0.0 to 5.8] | 0 [0.0 to 5.9] | 0 [0.0 to 6.0] | 0 [0.0 to 6.0] | 0 [0.0 to 5.7]
  Vomiting: Any | 0 [0.0 to 5.8] | 1.6 [0.0 to 8.8] | 3.3 [0.4 to 11.5] | 5.0 [1.0 to 13.9] | 1.6 [0.0 to 8.5]
  Vomiting: Mild | 0 [0.0 to 5.8] | 0 [0.0 to 5.9] | 3.3 [0.4 to 11.5] | 1.7 [0.0 to 8.9] | 1.6 [0.0 to 8.5]
  Vomiting: Moderate | 0 [0.0 to 5.8] | 1.6 [0.0 to 8.8] | 0 [0.0 to 6.0] | 3.3 [0.4 to 11.5] | 0 [0.0 to 5.7]
  Vomiting: Severe | 0 [0.0 to 5.8] | 0 [0.0 to 5.9] | 0 [0.0 to 6.0] | 0 [0.0 to 6.0] | 0 [0.0 to 5.7]
  Vomiting: Grade 4 | 0 [0.0 to 5.8] | 0 [0.0 to 5.9] | 0 [0.0 to 6.0] | 0 [0.0 to 6.0] | 0 [0.0 to 5.7]
  Diarrhea: Any | 12.9 [5.7 to 23.9] | 6.6 [1.8 to 15.9] | 16.7 [8.3 to 28.5] | 16.7 [8.3 to 28.5] | 12.7 [5.6 to 23.5]
  Diarrhea: Mild | 9.7 [3.6 to 19.9] | 6.6 [1.8 to 15.9] | 15.0 [7.1 to 26.6] | 13.3 [5.9 to 24.6] | 11.1 [4.6 to 21.6]
  Diarrhea: Moderate | 3.2 [0.4 to 11.2] | 0 [0.0 to 5.9] | 1.7 [0.0 to 8.9] | 3.3 [0.4 to 11.5] | 1.6 [0.0 to 8.5]
  Diarrhea: Severe | 0 [0.0 to 5.8] | 0 [0.0 to 5.9] | 0 [0.0 to 6.0] | 0 [0.0 to 6.0] | 0 [0.0 to 5.7]
  Diarrhea: Grade 4 | 0 [0.0 to 5.8] | 0 [0.0 to 5.9] | 0 [0.0 to 6.0] | 0 [0.0 to 6.0] | 0 [0.0 to 5.7]
  New or worsened muscle pain: Any | 25.8 [15.5 to 38.5] | 21.3 [11.9 to 33.7] | 45.0 [32.1 to 58.4] | 30.0 [18.8 to 43.2] | 27.0 [16.6 to 39.7]
  New or worsened muscle pain: Mild | 19.4 [10.4 to 31.4] | 8.2 [2.7 to 18.1] | 23.3 [13.4 to 36.0] | 11.7 [4.8 to 22.6] | 12.7 [5.6 to 23.5]
  New or worsened muscle pain: Moderate | 6.5 [1.8 to 15.7] | 11.5 [4.7 to 22.2] | 21.7 [12.1 to 34.2] | 18.3 [9.5 to 30.4] | 14.3 [6.7 to 25.4]
  New or worsened muscle pain: Severe | 0 [0.0 to 5.8] | 1.6 [0.0 to 8.8] | 0 [0.0 to 6.0] | 0 [0.0 to 6.0] | 0 [0.0 to 5.7]
  New or worsened muscle pain: Grade 4 | 0 [0.0 to 5.8] | 0 [0.0 to 5.9] | 0 [0.0 to 6.0] | 0 [0.0 to 6.0] | 0 [0.0 to 5.7]
  New or worsened joint pain: Any | 14.5 [6.9 to 25.8] | 14.8 [7.0 to 26.2] | 5.0 [1.0 to 13.9] | 13.3 [5.9 to 24.6] | 17.5 [9.1 to 29.1]
  New or worsened joint pain: Mild | 9.7 [3.6 to 19.9] | 6.6 [1.8 to 15.9] | 0 [0.0 to 6.0] | 3.3 [0.4 to 11.5] | 7.9 [2.6 to 17.6]
  New or worsened joint pain: Moderate | 4.8 [1.0 to 13.5] | 8.2 [2.7 to 18.1] | 5.0 [1.0 to 13.9] | 10.0 [3.8 to 20.5] | 9.5 [3.6 to 19.6]
  New or worsened joint pain: Severe | 0 [0.0 to 5.8] | 0 [0.0 to 5.9] | 0 [0.0 to 6.0] | 0 [0.0 to 6.0] | 0 [0.0 to 5.7]
  New or worsened joint pain: Grade 4 | 0 [0.0 to 5.8] | 0 [0.0 to 5.9] | 0 [0.0 to 6.0] | 0 [0.0 to 6.0] | 0 [0.0 to 5.7]

35. Primary Outcome: Cohort 4: Percentage of Participants With AEs From Study Vaccination Through 1 Month After Study Vaccination
Description: as for outcome 3
Time Frame: From study vaccination through 1 month after study vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 4: 18-55 Years (BNT162b2 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b5 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b6 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b7 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b7 Monovalent [OMI BA.4/ BA.5] 30 mcg)
Number analyzed (Participants) | 62 | 62 | 60 | 60 | 63
Percentage of participants | 8.1 [2.7 to 17.8] | 9.7 [3.6 to 19.9] | 1.7 [0.0 to 8.9] | 1.7 [0.0 to 8.9] | 1.6 [0.0 to 8.5]

36. Primary Outcome: Cohort 4: Percentage of Participants With SAEs From Study Vaccination Through 6 Months After Study Vaccination
Description: as for outcome 16
Time Frame: From study vaccination through 6 months after study vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 4: 18-55 Years (BNT162b2 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b5 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b6 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b7 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b7 Monovalent [OMI BA.4/ BA.5] 30 mcg)
Number analyzed (Participants) | 62 | 62 | 60 | 60 | 63
Percentage of participants | 1.6 [0.0 to 8.7] | 0 [0.0 to 5.8] | 0 [0.0 to 6.0] | 0 [0.0 to 6.0] | 0 [0.0 to 5.7]

37. Primary Outcome: Cohort 4: GMT of SARS-CoV-2 Omicron Strain (BA.4/BA.5) and Reference Strain NTs at Baseline- Participants With or Without Evidence of Infection
Description: as for outcome 6
Time Frame: At baseline (before study vaccination)
Population: EIP included all assigned/ randomized participants who received study intervention to which they were randomized/assigned, had at least 1 valid and determinate immunogenicity result from blood sample collected within 28-42 days post the vaccination and had no other important protocol deviations. Analysis was performed in participants with or without evidence of infection up to 1 month post study vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 4: 18-55 Years (BNT162b2 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b5 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b6 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b7 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b7 Monovalent [OMI BA.4/ BA.5] 30 mcg)
Number analyzed (Participants) | 61 | 61 | 57 | 56 | 61
Titer
  Omicron BA.4/BA.5 | 1332.5 [909.2 to 1953.0] | 1313.6 [922.6 to 1870.2] | 1352.0 [876.0 to 2086.8] | 1320.1 [869.8 to 2003.6] | 1203.9 [796.5 to 1819.6]
  Reference strain | 3445.5 [2465.4 to 4815.3] | 4907.1 [3753.0 to 6416.1] | 4613.6 [3474.3 to 6126.4] | 4395.7 [3244.1 to 5956.3] | 4318.6 [3196.1 to 5835.2]

38. Primary Outcome: Cohort 4: GMT of SARS-CoV-2 Omicron Strain (BA.4/BA.5) and Reference Strain NTs at 1 Month After Study Vaccination- Participants With or Without Evidence of Infection
Description: as for outcome 6
Time Frame: 1 month after the study vaccination
Population: as for outcome 37
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 4: 18-55 Years (BNT162b2 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b5 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b6 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b7 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b7 Monovalent [OMI BA.4/ BA.5] 30 mcg)
Number analyzed (Participants) | 61 | 61 | 57 | 56 | 61
Titer
  Omicron BA.4/BA.5 | 4850.5 [3677.1 to 6398.3] | 4854.3 [3713.9 to 6344.9] | 4944.6 [3620.3 to 6753.1] | 5180.6 [3724.6 to 7205.8] | 5455.6 [4214.2 to 7062.8]
  Reference strain | 10455.0 [8150.7 to 13410.8] | 11360.0 [9408.3 to 13716.6] | 10840.2 [8475.3 to 13865.0] | 12303.8 [9728.6 to 15560.5] | 11164.3 [8729.0 to 14279.0]

39. Primary Outcome: Cohort 4: GMFR of SARS-CoV-2 Omicron Strain (BA.4/BA.5) and Reference Strain- NTs From Before the Study Vaccination to 1 Month After the Study Vaccination- Participants With or Without Evidence of Infection
Description: as for outcome 10
Time Frame: From before the study vaccination to 1 month after study vaccination
Population: as for outcome 37
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Cohort 4: 18-55 Years (BNT162b2 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b5 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b6 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b7 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b7 Monovalent [OMI BA.4/ BA.5] 30 mcg)
Number analyzed (Participants) | 61 | 61 | 57 | 56 | 61
Fold rise
  Omicron BA.4/BA.5 | 3.6 [2.7 to 4.8] | 3.7 [2.7 to 5.0] | 3.7 [2.8 to 4.7] | 3.9 [2.9 to 5.3] | 4.5 [3.3 to 6.2]
  Reference strain | 3.0 [2.3 to 4.0] | 2.3 [1.8 to 3.0] | 2.3 [1.9 to 2.8] | 2.8 [2.1 to 3.7] | 2.6 [2.1 to 3.2]

40. Primary Outcome: Cohort 4: Percentage of Participants With Seroresponse to SARS-CoV-2 Omicron Strain (BA.4/BA.5) and Reference Strain- NTs at 1 Month After Study Vaccination- Participants With or Without Evidence of Infection
Description: as for outcome 11
Time Frame: 1 month after study vaccination
Population: as for outcome 37
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 4: 18-55 Years (BNT162b2 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b5 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b6 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b7 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b7 Monovalent [OMI BA.4/ BA.5] 30 mcg)
Number analyzed (Participants) | 61 | 61 | 57 | 56 | 61
Percentage of participants
  Omicron BA.4/BA.5 | 42.6 [30.0 to 55.9] | 41.0 [28.6 to 54.3] | 42.1 [29.1 to 55.9] | 39.3 [26.5 to 53.2] | 44.3 [31.5 to 57.6]
  Reference strain | 37.7 [25.6 to 51.0] | 27.9 [17.1 to 40.8] | 22.8 [12.7 to 35.8] | 26.8 [15.8 to 40.3] | 29.5 [18.5 to 42.6]

ADVERSE EVENTS:
Time Frame: Local reactions and systemic events: From Day 1 to Day 7 after study vaccination; AE: From study vaccination on Day 1 through 1 month after study vaccination, SAE and Death: From study vaccination on Day 1 through 6 months after study vaccination
Description: Same event may appear as non-SAE and SAE, what is presented are distinct. Event may be categorized as serious in 1 participant and non-serious in other, or participant may experience both SAE and non-SAE. Safety population: all participants who received study intervention and where appropriate informed consent was obtained. Per analysis planned, data is summarized & combined for Cohort 2/ Cohort 3 30 mcg groups per age category. MedDRA for Cohort1/Cohort 4: v27.0; for Cohort 2/Cohort 3: v26.0.
Arm/Group | Cohort 1: 18-55 Years (BNT162b5 Bivalent [WT/ OMI BA.2] 30 mcg) | Cohort 1: 18-55 Years (BNT162b2 Bivalent [WT/ OMI BA.1] 30 mcg) | Cohort 2 (Group 1): 12-17 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 30 mcg) | Cohort 2 (Group 2) + Cohort 3 (Group 1): 18-55 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 30 mcg) | Cohort 2 (Group 3): 18-55 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 60 mcg) | Cohort 2 (Group 4) + Cohort 3 (Group 2): >55 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 30 mcg) | Cohort 2 (Group 5): >55 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 60 mcg) | Cohort 4: 18-55 Years (BNT162b2 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b5 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b6 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b7 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) | Cohort 4: 18-55 Years (BNT162b7 Monovalent [OMI BA.4/ BA.5] 30 mcg)
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/102 | 0/107 | 0/313 | 0/110 | 1/306 | 0/102 | 0/62 | 0/62 | 0/60 | 0/60 | 0/63
Serious Adverse Events (participants affected / at risk) | 1/104 | 2/102 | 1/107 | 2/313 | 1/110 | 10/306 | 0/102 | 1/62 | 0/62 | 0/60 | 0/60 | 0/63
Other Adverse Events (participants affected / at risk) | 97/104 | 91/102 | 96/107 | 269/313 | 106/110 | 210/306 | 82/102 | 55/62 | 56/62 | 52/60 | 53/60 | 56/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: 18-55 Years (BNT162b5 Bivalent [WT/ OMI BA.2] 30 mcg) (N=104) | Cohort 1: 18-55 Years (BNT162b2 Bivalent [WT/ OMI BA.1] 30 mcg) (N=102) | Cohort 2 (Group 1): 12-17 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 30 mcg) (N=107) | Cohort 2 (Group 2) + Cohort 3 (Group 1): 18-55 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 30 mcg) (N=313) | Cohort 2 (Group 3): 18-55 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 60 mcg) (N=110) | Cohort 2 (Group 4) + Cohort 3 (Group 2): >55 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 30 mcg) (N=306) | Cohort 2 (Group 5): >55 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 60 mcg) (N=102) | Cohort 4: 18-55 Years (BNT162b2 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) (N=62) | Cohort 4: 18-55 Years (BNT162b5 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) (N=62) | Cohort 4: 18-55 Years (BNT162b6 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) (N=60) | Cohort 4: 18-55 Years (BNT162b7 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) (N=60) | Cohort 4: 18-55 Years (BNT162b7 Monovalent [OMI BA.4/ BA.5] 30 mcg) (N=63)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular germ cell cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: 18-55 Years (BNT162b5 Bivalent [WT/ OMI BA.2] 30 mcg) (N=104) | Cohort 1: 18-55 Years (BNT162b2 Bivalent [WT/ OMI BA.1] 30 mcg) (N=102) | Cohort 2 (Group 1): 12-17 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 30 mcg) (N=107) | Cohort 2 (Group 2) + Cohort 3 (Group 1): 18-55 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 30 mcg) (N=313) | Cohort 2 (Group 3): 18-55 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 60 mcg) (N=110) | Cohort 2 (Group 4) + Cohort 3 (Group 2): >55 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 30 mcg) (N=306) | Cohort 2 (Group 5): >55 Years (BNT162b2 Bivalent [WT/ OMI BA.4/ BA.5] 60 mcg) (N=102) | Cohort 4: 18-55 Years (BNT162b2 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) (N=62) | Cohort 4: 18-55 Years (BNT162b5 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) (N=62) | Cohort 4: 18-55 Years (BNT162b6 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) (N=60) | Cohort 4: 18-55 Years (BNT162b7 Bivalent [Original/ OMI BA.4/ BA.5] 30 mcg) (N=60) | Cohort 4: 18-55 Years (BNT162b7 Monovalent [OMI BA.4/ BA.5] 30 mcg) (N=63)
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 19 (19) | 18 (18) | 13 (13) | 46 (46) | 27 (27) | 36 (36) | 15 (15) | 9 (9) | 9 (9) | 3 (3) | 8 (8) | 11 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bell's palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (CHILLS) (General disorders) | 22 (22) | 20 (20) | 25 (25) | 68 (68) | 30 (30) | 36 (36) | 23 (23) | 14 (14) | 11 (11) | 17 (17) | 8 (8) | 12 (12)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (DIARRHEA) (Gastrointestinal disorders) | 15 (15) | 20 (20) | 7 (7) | 33 (33) | 14 (14) | 28 (28) | 7 (7) | 8 (8) | 4 (4) | 10 (10) | 10 (10) | 8 (8)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Fatigue (FATIGUE) (General disorders) | 76 (76) | 64 (64) | 72 (72) | 189 (189) | 76 (76) | 115 (115) | 54 (54) | 38 (38) | 39 (39) | 44 (44) | 39 (39) | 34 (34)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (HEADACHE) (Nervous system disorders) | 55 (55) | 47 (47) | 54 (54) | 144 (144) | 50 (50) | 92 (92) | 36 (36) | 37 (37) | 22 (22) | 25 (25) | 28 (28) | 25 (25)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (REDNESS) (General disorders) | 6 (6) | 6 (6) | 6 (6) | 20 (20) | 12 (12) | 11 (11) | 7 (7) | 3 (3) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 3 (3)
Injection site pain (PAIN) (General disorders) | 86 (86) | 83 (83) | 75 (75) | 235 (235) | 103 (103) | 171 (171) | 71 (71) | 52 (52) | 54 (54) | 45 (45) | 46 (46) | 52 (52)
Injection site swelling (SWELLING) (General disorders) | 11 (11) | 11 (11) | 8 (8) | 22 (22) | 17 (17) | 8 (8) | 9 (9) | 1 (1) | 2 (2) | 4 (4) | 2 (2) | 2 (2)
Joint abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 37 (37) | 39 (39) | 28 (28) | 94 (94) | 46 (46) | 54 (54) | 23 (23) | 16 (16) | 13 (13) | 27 (27) | 17 (17) | 17 (17)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (FEVER) (General disorders) | 2 (2) | 6 (6) | 10 (10) | 15 (15) | 13 (13) | 13 (13) | 14 (14) | 4 (4) | 4 (4) | 6 (6) | 3 (3) | 6 (6)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (VOMITING) (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 6 (6) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/38/NCT05472038/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-04): https://cdn.clinicaltrials.gov/large-docs/38/NCT05472038/SAP_001.pdf